## STATISTICAL ANALYSIS PLAN

Study Title: A Phase 2 Study of Tarloxotinib in Patients with Select

Gene Alterations and Non-Small Cell Lung Cancer or

Other Advanced Solid Tumors

**Study Number:** RAIN-701

**Investigational Drug:** Tarloxotinib bromide

**Indication:** Treatment of Non-Small Cell Lung Cancer or Other

**Advanced Solid Tumors** 

**Investigators:** Multicenter

**IND Number:** 112290

**Sponsor:** Rain Therapeutics Inc.

8000 Jarvis Ave Suite 204

Newark, CA, 94560

**Plan Version:** 1.0, 14 October 2022

Plan Prepared by: Inka Leprince, MS

Statistical Consultant

PharmaStat, LLC

## CONFIDENTIAL

This document is confidential and property of Rain Therapeutics Inc. It may not be copied or provided to any other party without the express written consent of Rain Therapeutics Inc.

©2022 Rain Therapeutics Inc.

## STATISTICAL ANALYSIS PLAN

## **RAIN-701**

A Phase 2 Study of Tarloxotinib in Patients with Select Gene Alterations and Non-Small Cell Lung Cancer or Other Advanced Solid Tumors

| Plan Version | n: 1.0, 14 October 2022 | |
|---|---|---|
| Plan version | reviewed: 14 October 2022 | |
| Signature Pa | ageDocuSigned by: | |
| Author: | / nla La | |
| | Inka Leprince, MS Statistician and Data Analyst PharmaStat, LLC | Date |
| Reviewer: | DocuSigned by: ( | |
| | Lucio Tozzi SVP, Head of Clinical Operations Rain Therapeutics Inc. | Date |
| Reviewer: | Robert C Double | |
| | Robert & Doebele, MD, PhD President and Chief Scientific Officer Rain Therapeutics Inc. | Date |
| Reviewer: | DocuSigned by: Fug Xu 0E8D70E3F53B44F | |
| | Feng Xu VP, Biometrics Rain Therapeutics Inc. | Date |

## **Table of Contents**

| 1 | REVISION HISTORY | 9 |
|-------|---------------------------------------------------|----|
| 2 | RELATED DOCUMENTS: PROTOCOL AND CASE REPORT FORMS | 9 |
| 3 | COMMITMENT TO GOOD STATISTICAL PRACTICE | 9 |
| 3.1 | Definition of Good Statistical Practice | 9 |
| 3.2 | Use of Standards | 9 |
| 4 | PURPOSE OF THE ANALYSIS PLAN | 10 |
| 5 | STUDY OBJECTIVE | 11 |
| 5.1 | Efficacy Objectives and Endpoints | 11 |
| 5.1.1 | Primary Efficacy | 11 |
| 5.1.2 | Secondary Efficacy | 11 |
| 5.1.3 | Exploratory Efficacy | 12 |
| 5.2 | Safety Objective | 12 |
| 6 | STUDY DESIGN | 12 |
| 6.1 | Overall Study Design | 12 |
| 6.2 | Study Medication | 14 |
| 6.2.1 | Tarloxotinib | 14 |
| 6.2.2 | Potassium Supplementation | 14 |
| 6.2.3 | Premedication | 15 |
| 6.3 | Assessments | 15 |
| 6.3.1 | Efficacy Assessments | 15 |
| 6.3.2 | Safety Assessments | 16 |
| 6.3.3 | Pharmacokinetic Measurements | 17 |
| 6.3.4 | Tumor Tissue | 17 |
| 6.3.5 | Biomarker Analysis | 17 |
| 7 | SAMPLE SIZE AND POWER | 20 |
| 8 | ANALYSIS SETS | 20 |
| 8.1 | Intent-To-Treat Analysis Set | 20 |
| 8.2 | Primary Analysis Set | 20 |
| 9 | GENERAL CONSIDERATIONS | 20 |
| 9.1 | Presentation of Summary Statistics | 20 |
| 9.2 | Definitions and Derived Variables | 21 |
| 9.2.1 | Screened and Enrolled Subjects | 21 |
| 9.2.2 | Study Day | 21 |
| 9.2.3 | End of Study Treatment Definition | 22 |
| 9.2.4 | End of Study Definition | 22 |
| 9.2.5 | Date Last Known Alive | 22 |

# Version 1.0, 14 October 2022

| 101111 / 0 | Version 1.0, 14 Cetober 2 | 022 |
|------------|-------------------------------------------------------|-----|
| 9.2.6 | Age | 22 |
| 9.2.7 | Body Mass Index | |
| 9.2.8 | Baseline Values | 22 |
| 9.2.9 | Sum of Target Lesions | 22 |
| 9.2.10 | Evaluable Subjects | 23 |
| 9.2.11 | RECIST Response Assessment | 23 |
| 9.2.12 | Duration of Response | 24 |
| 9.2.13 | Disease Control Rate | 24 |
| 9.2.14 | Progression-Free Survival | 25 |
| 9.2.15 | Overall Survival | 25 |
| 9.2.16 | Study Drug Exposure Variables | 25 |
| 9.2.17 | Prior, Concomitant and Post treatment Medications | |
| 9.2.18 | Adverse Events | 26 |
| 9.3 | Analysis Windows | 28 |
| 10 | STATISTICAL AND ANALYSIS ISSUES | 29 |
| 10.1 | Adjustments for Covariates | 29 |
| 10.2 | Handling Dropouts or Missing Data | 29 |
| 10.2.1 | Handling of Laboratory Data | |
| 10.2.2 | Handling of Safety Data | |
| 10.3 | Multicenter Considerations | |
| 10.4 | Multiple Comparisons, Multiplicity | 31 |
| 10.5 | Active-Control Studies | 31 |
| 10.6 | Examination of Subgroups | 31 |
| 11 | STUDY SUBJECTS | 31 |
| 11.1 | Subject Enrollment and Disposition | 31 |
| 11.1.1 | Enrolled Subjects | 31 |
| 11.2 | Protocol Deviations | 32 |
| 11.3 | Demographics and Baseline Characteristics | 32 |
| 11.3.1 | Key Baseline Demographics | 32 |
| 11.4 | Medical History | 32 |
| 12 | STUDY DRUG AND OTHER MEDICATIONS | 33 |
| 12.1 | Exposure to Study Drug and Study Treatment Compliance | 33 |
| 12.2 | Prior and Concomitant Medications | 33 |
| 13 | EFFICACY ANALYSES | 34 |
| 13.1 | Primary Analysis | 34 |
| 13.2 | Primary Efficacy | 34 |
| 13.3 | Secondary Efficacy | 34 |

| Rain The | erapeutics Inc. 01 SAP Version 1.0, 14 Octob | 2022 |
|---|---|---|
| KAIN-/ | JI SAF VEISIOII 1.0, 14 Octob | <u> </u> |
| 13.3.1 | Duration of Response | 35 |
| 13.3.2 | Survival Reporting | 35 |
| 13.4 | Exploratory Objectives | 35 |
| 13.5 | Subgroup Analyses | 35 |
| 14 | SAFETY ANALYSES | 36 |
| 14.1 | Adverse Events | 36 |
| 14.1.1 | Overall Summary of TEAEs | 36 |
| 14.1.2 | Summary of TEAEs by System Organ Class and Preferred Term | 37 |
| 14.1.3 | Summary of TEAEs by Preferred Term | 37 |
| 14.2 | Clinical Laboratory Evaluation | 37 |
| 14.3 | Vital Signs | 38 |
| 14.4 | 12-Lead Electrocardiogram | |
| 15 | CHANGES RELATIVE TO THE PROTOCOL-SPECIFIED ANALYSIS | 40 |
| 16 | References | 42 |
| 17 | Appendix A: Local Laboratory Units and Reference Ranges by Site and Parameter | 43 |
| 18 | Appendix B: | 58 |
| <b>List of T</b> : Table 1 | ables RAIN-701 Number of Subjects by Cohort | 12 |
| Table 2 | Study RAIN-701 Protocol Schedule Events (Protocol [Amendment 3] 24 Octo 2020) | ober |
| Table 3 | Response Evaluation Criteria in Solid Tumours Guidelines | 23 |
| Table 4 | Censoring Rules for Progression-Free Survival | 24 |
| Table 5 | Severity Grading Guideline for Adverse Events | 27 |
| Table 6 | Visit Analysis Windows (Clinic visits only) | |
| Table 7 | Clinical Laboratory Parameters | |
| Table 8 | Site 101 Units and Reference Ranges by Parameter | |
| Table 9 | Site 102 Units and Reference Ranges by Parameter | |
| Table 10 | Site 103 Units and Reference Ranges by Parameter | |
| Table 11 | Site 104 Units and Reference Ranges by Parameter | |
| Table 12 | Site 105 Units and Reference Ranges by Parameter | |
| Table 13 | Site 107 Units and Reference Ranges by Parameter | |
| Table 14 | | |
| | Site 111 Units and Reference Ranges by Parameter | |
| | <i>O</i> | |

## 

| | List of Abbreviations and Definition of Terms |
|---|---|
| Abbreviation | Description |
| ADaM | analysis data model |
| AE | adverse event |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| ATC | Anatomical / Therapeutic / Chemical |
| BOR | best overall response |
| CI | confidence interval |
| CDISC | Clinical Data Interchange Standards Consortium |
| CM | concomitant medication |
| CR | complete response |
| CSR | clinical study report |
| CT | computed tomography |
| ctDNA | circulating tumor deoxyribonucleic acids |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DCR | disease control rate |
| DOR | duration of response |
| ECG | electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| EGFR | epidermal growth factor receptor |
| EOI | End of infusion |
| EOT | End-of-Treatment Visit |
| ERBB2 | v-erb-b2 avian erythroblastic leukemia viral oncogene homolog 2 |
| ERBB4 | erb-b2 Receptor tyrosine kinase 4 |
| FDA | Food and Drug Administration |
| HER | human epidermal growth factor receptor |
| HR | heart rate |
| ICH | International Council for Harmonisation |
| IV | intravenous |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | magnetic resonance imaging |
| NCI | National Cancer Institute |
| NRG1 | neuregulin 1 |
| NSCLC | non-small cell lung cancer |
| ORR | objective response rate |

## Rain Therapeutics Inc.

RAIN-701 SAP

Version 1.0, 14 October 2022

| Abbreviation | Description |
|---|---|
| OS | overall survival |
| PAS | Primary analysis set |
| PD | progressive disease |
| PET | positron emissions tomography |
| PFS | progression-free survival |
| PK | pharmacokinetic |
| PO | oral |
| PR | partial response |
| QTc | corrected QT interval |
| QTcF | corrected QTc interval as calculated according to Fridericia's formula |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | stable disease (tumor response) |
| SD | standard deviation (statistics) |
| SOC | system organ class |
| STEAP4 | six transmembrane epithelial antigen of the prostate, family member 4 |
| TEAE | treatment-emergent adverse event |
| TLF | tables, listings, and figures |
| WHO | World Health Organization |
| WOCBP | women of childbearing potential |


#### 1 REVISION HISTORY

| Version | Date | Document<br>Owner | Revision Summary |
|---------|--------------------|-------------------|------------------|
| 1.0 | 14 October<br>2022 | Inka Leprince | Initial version |

#### 2 RELATED DOCUMENTS: PROTOCOL AND CASE REPORT FORMS

| Version | Date |
|--------------------------|-----------|
| Initial Protocol | 14Dec2018 |
| Protocol (Amendment 1) | 06Mar2019 |
| Protocol (Amendment 2) | 17Jun2019 |
| Protocol (Amendment 2.1) | 11Nov2019 |
| Protocol (Amendment 3) | 24Oct2020 |
| Case Report Forms | 22Mar2019 |

#### 3 COMMITMENT TO GOOD STATISTICAL PRACTICE

## 3.1 Definition of Good Statistical Practice

The International Council for Harmonisation Guideline on Statistical Principles for Clinical Trials (ICH E9) implicitly defines good statistical practice. Good statistical practice includes both appropriate statistical designs to minimize bias and maximize precision of analysis plus operational excellence to assure credibility of results. The scientific design associated with any clinical trial is found in the protocol and a more detailed, pre-specified statistical analysis plan such as this one presents the final statistical methods.

We interpret the operational side of good statistical practice as a transparent, reproducible, and validated approach to acquiring and analyzing clinical trial data. Reproducible research depends upon process transparency and also provides auditability of the statistical analysis. Analysis transparency requires that a navigable electronic process chain exists from defining the objective of the analysis to creating the results.

#### 3.2 Use of Standards

Data standards are foundational for creating an environment where tools can be leveraged at different points in the analysis process. Data standards for clinical development of drugs have been defined and are maturing under various initiatives through the Clinical Data Interchange


Standards Consortium (CDISC). RAIN Therapeutics uses raw, source data sets and Analysis Data Model (ADaM) statistical analysis files for producing analysis results. Other applicable standards include regulatory guidance from the Food and Drug Administration (FDA) and ICH:

- ICH Guideline on the Structure and Content of Clinical Study Reports (ICH E3)
- ICH Guideline for Good Clinical Practice (ICH E6)

#### 4 PURPOSE OF THE ANALYSIS PLAN

This statistical analysis plan (SAP) pre-specifies the statistical analysis methods for supporting the completion of the abbreviated clinical study report (CSR) of Study RAIN-701 for investigational product tarloxotinib, a novel drug candidate designed to treat subjects with advanced solid tumors with qualifying genetic mutations and/or fusions. The study intended to enroll up to 215 subjects across 5 cohorts but was discontinued early on the basis of a business decision made by the sponsor. At the time of the database lock for RAIN-701 (23 April 2021), 41 subjects were enrolled. This SAP will be used to conduct a comprehensive safety analysis and summarize the available efficacy data collected during the study. The primary, secondary, and efficacy analyses planned in the protocol may not be appropriate or possible based on the available data. The planned analyses identified in this SAP may be included in future manuscripts.

The analysis methods described in this plan are considered *a posterior*, in that they have been defined after the clinical database lock. Exploratory analyses that are not defined in this SAP may be performed to support the clinical development program. Any post-hoc or unplanned analyses that are performed for the CSR, but not defined in this SAP, will be documented in the CSR. Changes from the planned analyses stated in the study protocol are described in Section 15. Should the SAP and the protocol be inconsistent with respect to any further planned analyses, the language of the SAP is governing.


#### 5 STUDY OBJECTIVE

This study was planned to evaluate the safety and efficacy of tarloxotinib 150 mg/m² as a weekly 1-hour intravenous (IV) infusion of up to 40 weeks when administered to subjects with non-small cell lung cancer (NSCLC) whose tumors harbor either an epidermal growth factor receptor (EGFR) exon 20 insertion or a human epidermal growth factor receptor 2 (HER2)-activating mutation (including exon insertions).

## 5.1 Efficacy Objectives and Endpoints

The primary, secondary, and efficacy analyses planned in the protocol may not be appropriate or possible based on the available data. Additionally, efficacy analyses are unlikely to be significant because the sample size is small and the analyses will be underpowered. In place of formal efficacy analyses, selected efficacy endpoints will be summarized descriptively.

## 5.1.1 Primary Efficacy

The analysis of the primary objective as outlined in the study protocol will not be performed for the abbreviated CSR, but will instead be summarized descriptively and listed where possible. The primary objective of this study was the evaluation of the objective response rate (ORR), based on subjects who had complete response or partial response, of tarloxotinib according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

## 5.1.2 Secondary Efficacy

The analyses of the secondary objectives as outlined in the study protocol will not be performed for the abbreviated CSR, but will instead be summarized descriptively and listed where possible. Secondary objectives include evaluation of the antitumor effect of tarloxotinib on: best overall response (BOR), duration of response (DOR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS) as measured from the date of first study drug dose to the date of death by any cause. Additional secondary efficacy endpoints such as the exploration of pharmacokinetics of tarloxotinib and tarloxotinib-E; and the determination of whether there is

an association between plasma exposure to tarloxotinib and effects on cardiac repolarization will not be performed because of the limited data basis.

## 5.1.3 Exploratory Efficacy

The analyses of the exploratory objectives as outlined in the study protocol will not be performed for the abbreviated CSR because of the limited data basis. Exploratory objectives are described in Protocol Section 4.2.3.

## 5.2 Safety Objective

The safety objective of the study is to evaluate the safety of tarloxotinib subjects with NSCLC using safety assessments described in Section 6.3.2. Safety endpoints include the incidence of treatment-emergent adverse events (TEAEs); changes in clinical laboratory parameters (hematology, serum chemistry, and urinalysis), vital signs, and electrocardiogram (ECG) parameters; physical examination results; and use of concomitant medications (CMs).

#### 6 STUDY DESIGN

#### 6.1 Overall Study Design

This was a Phase 2 multicenter, open-label study to evaluate the antitumor effect of tarloxotinib in subjects with NSCLC whose tumors harbors either an EGFR exon 20 insertion or a HER2-activating mutation (including exon 20 insertions) or subjects with advanced solid tumors expressing NRG1/HER-family gene fusions or a HER2-activating. All subjects have received at least 1 prior platinum-based chemotherapy-containing regimen in the advanced/metastatic setting (Cohorts A, B, and B1) or standard of care for cancer (Cohorts C and D). Cohorts B1 and D were not be pursued at the discretion of the Sponsor.

Table 1 RAIN-701 Number of Subjects by Cohort

| Cohort | Description | Planned<br>N | Enrolled<br>N |
|---|---|---|---|
| A: | Subjects with advanced NSCLC harboring an EGFR exon 20 insertion mutation o At least 1 prior platinum-based chemotherapy-containing regimen | 43 | 11 |
| B: | Subjects with advanced NSCLC with a HER2 activating mutation | 43 | 22 |


| | Subjects who have received at least 1 prior platinum-based chemotherapy-containing regimen | | |
|---|---|---|---|
| B1* | <ul> <li>Subjects with advanced NSCLC harboring a HER2-activating mutation</li> <li>Subjects who have received at least 1 platinum-based chemotherapy-containing regimen</li> <li>Subjects who have received prior HER2-directed therapy</li> </ul> | 43 | 0 |
| C: | <ul> <li>Subjects with advanced solid tumors who have failed standard therapies appropriate for their tumor type and stage of disease, or, in the opinion of the Investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard-of-care therapy</li> <li>Subjects with tumors harboring an NRG1 gene fusion, EGFR gene fusion, EGFR kinase domain duplication, ERBB2 gene fusion, or ERBB4 gene fusion</li> </ul> | 43 | 8 |
| D*: | <ul> <li>Subjects with advanced solid tumors who have failed all standard therapies appropriate for their tumor type and stage of disease, or, in the opinion of the Investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard-of-care therapy</li> <li>Subjects with tumors (excluding NSCLC) harboring a HER2-activating mutation</li> </ul> | 43 | 0 |
| Total | | 215 | 41 |

Approximately 248 subjects were planned for enrollment on the study to yield 215 evaluable subjects, 43 subjects per cohort. A total of 41 subjects were enrolled in cohorts A, B and C. No subjects were enrolled on cohorts C and D. All cohorts used a Simon's 2-stage design. In the first stage, 21 subjects were accrued. If more than 3 subjects in a cohort had a partial or complete response, up to 22 additional subjects could have been enrolled to the cohort, for up to a total of 43 subjects per cohort. However, if there were 3 or fewer responses among these 21 subjects, the cohort would be stopped based on futility.

Subjects received taroxontinib 150 mg/m<sup>2</sup> administered as a weekly 1-hour IV infusion on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression or unacceptable toxicity (e.g., hepatotoxicity meeting Hy's law criteria or serious arrhythmias of ventricular origin).

<sup>\*</sup> Cohorts B1 and/or D were not pursued, at the discretion of the Sponsor

Subjects were expected to receive up to 10 cycles of treatment. The total study duration was estimated to be 36 months, including approximately 24 months for accrual and approximately 12 months for follow-up after the last subject was enrolled. Upon completion of the end of treatment visit, subjects returned to the clinic within 30 days following their last dose for a Follow-up visit. Clinical visits during the Treatment Period and Follow-up Period included efficacy, biomarkers, safety, and pharmacokinetic (PK) assessments. Figure 1 depicts study visits from Screening Period to Follow-up Period. The maximum duration of Study RAIN-701 per subject was expected to be up to 338 days (i.e., a maximum of 28-day Screening Period, a Treatment Period consisting of a maximum of ten 28-day treatment cycles, and a 30-day safety Follow-up Period). Assessments and procedures for evaluation of safety, efficacy, PK, and biomarkers were conducted per the protocol-specified schedule (see Table 2).

Figure 1 Schema of Study RAIN-701



Days 1, 8, 15, and 22 of every 28-day cycle

#### **6.2** Study Medication

#### 6.2.1 Tarloxotinib

Tarloxotinib 150 mg/m² was administered as a 1-hour IV infusion weekly until progressive disease (PD) or unacceptable toxicity. Tarloxotinib was administered on Day 1, Day 8, Day 15, and Day 22 of every 28-day cycle. All infusions after Cycle 1 Day 1 were administered 7 days  $\pm$  1 day after the prior infusion.

## **6.2.2** Potassium Supplementation

Serum electrolytes (including potassium) were checked prior to each tarloxotinib infusion. Subjects with a pre-infusion serum potassium of < 3.5 mEq/L received potassium replacement

<sup>&</sup>lt;sup>2</sup> Every 8 weeks( $\pm$  5 days) from Cycle 1 Day 1

per institutional policy (IV and/or oral [PO]) and have the scheduled tarloxotinib infusion delayed at least 24 hours and potassium levels rechecked within 1 hour prior to the rescheduled infusion. All subjects with a pre-infusion serum potassium levels  $\geq 3.5$  mEq/L and  $\leq 5.0$  mEq/L were supplemented daily with 40 mEq/L of potassium replacement per institutional policy (IV and/or PO).

#### 6.2.3 Premedication

All subjects may have received steroid or anti-emetics premedication prior to tarloxotinib infusions. The premedication regimen was determined by the Investigator and may be adjusted at subsequent infusions based on the signs and symptoms observed during or after prior infusions.

#### 6.3 Assessments

Table 2 shows the schedule of events for the study.

## **6.3.1** Efficacy Assessments

Tumor assessment and imaging was performed according to institutional practice and included computerized tomography (CT) or magnetic resonance imaging (MRI) of the chest and abdomen, brain scan, and bone scan at baseline. The baseline radiographic tumor assessment was required within 28 days prior to the first dose of tarloxotinib, at the Screening assessment. Brain and bone scans did not need to be repeated for subjects with no brain or bone metastases at baseline. Recently completed negative positron emissions tomography (PET) scans could be substituted for baseline bone scans. Subsequent radiographic tumor assessments were every 8 weeks (± 5 days) with respect to Cycle 1 Day 1 (e.g., Cycle 3 Day 1, Cycle 5 Day 1, etc.), until unequivocal PD was documented. The same imaging modality used for baseline imaging (i.e., CT or MRI) was used for subsequent tumor assessments in each subject. In accordance with RECIST v1.1, response (partial response [PR] and complete response [CR]) was confirmed by a second tumor assessment at least 4 weeks after the initial observed response. The scheduling of subsequent tumor assessments may have been adjusted based on the date of the most recent imaging.

## **6.3.2** Safety Assessments

The objective of the safety assessments was to evaluate the safety and tolerability of tarloxotinib in this population, including to determine whether there is an association between plasma exposure to tarloxotinib and effects on cardiac repolarization. Safety was assessed by repeated clinical evaluations including adverse events (AEs), suspected adverse reactions, unexpected events, serious AEs (SAEs), serious unexpected suspected adverse reactions, vital signs, physical examination, ECGs, clinical laboratory tests (serum chemistry, hematology, and urinalysis).

## 6.3.2.1 Adverse Events

Investigators collected information related to AEs throughout this clinical trial. All AEs occurring in all subjects were collected following exposure to study treatment (treatment emergent) until approximately 30 days after the last study treatment.

## 6.3.2.2 Vital Signs

Vital signs were obtained at each visit and prior to and following the start of each tarloxotinib infusion. Vital signs measured include: blood pressure (systolic and diastolic; mmHg); heart rate (beats per minute); body temperature (°C); respiration rate (breaths per minute); and weight (kg).

## **6.3.2.3** Physical Examinations

Complete physical examinations, including a review of all body systems, was performed at the Screening, Day 1 of all cycles, and the end of treatment (EOT) visits as shown in Table 2. Clinically significant findings observed during physical examination were reported as medical history (pre-treatment) or AEs (post-treatment).

## 6.3.2.4 Electrocardiograms

All 12-lead ECG tracings were performed once at the following visits: Screening, EOT, and Safety Follow-up. During Cycle 1, ECGs were performed at five time points (preinfusion, end of infusion [EOI], 1 hour after EOI, 2 hours after EOI, 3 hours after EOI, 4 hours after EOI), and hourly thereafter as needed. After Cycle 1, all treatment visits have ECGs performed at a minimum of three time points (preinfusion, 2 hours after EOI, 4 hours after EOI) and hourly thereafter as needed, as shown in Table 2.

#### **6.3.3** Pharmacokinetic Measurements

Blood samples for tarloxotinib and tarloxotinib-E plasma concentrations were collected prior to and following tarloxotinib infusion on Cycle 1 Day 1 and Cycle 2 Day 1. Serum potassium samples were also collected after the infusion. All blood samples may be collected within the 5 or 10 minutes (see Table 2) prior to or following the protocol-specified time point.

Plasma samples were collected for evaluation of the pharmacokinetics of tarloxotinib and tarloxotinib-E in tumor tissue. Plasma sample were collected at approximately at pre-infusion, EOI, 3 hours after EOI, and 7 hours after EOT (Cycle 1 Day 1 only) for measurement of tarloxotinib and tarloxotinib-E concentrations at each Cycle 1 Day 1 and Cycle 2 Day 1 visits as indicated in Table 2. An optional tumor biopsy may have been conducted at Cycle 1 Day 15.

#### **6.3.4** Tumor Tissue

All subjects had tumor tissue collected at baseline. Tumor samples obtained during screening may have also been used to determine levels of the reductase, six transmembrane epithelial antigen of the prostate, family member 4 (STEAP4). In addition to the above-mentioned tumor sample, an optional tumor tissue sample for measurement of the active metabolite (tarloxotinib-E) and tarloxotinib may have been collected from consenting subjects on Cycle 1 Day 15 after infusion along with a blood sample for PK. If the biopsy (and associated PK sample) was not able to be performed on the Cycle 1 Day 15 visit, it should have been collected within the 24 hours after the tarloxotinib infusion or after another infusion day.

## 6.3.5 Biomarker Analysis

Blood samples were collected for biomarker assessment (e.g., circulating tumor deoxyribonucleic acid [ctDNA]) at the Cycle 1 Day 1, Cycle 2 Day 2, and End of Treatment visits. Biomarker assessment may include ctDNA mutation analysis and evaluation of the concordance of EGFR and HER2 mutation identification between blood and tumor tissue.


Rain Therapeutics Inc. RAIN-701 SAP Study RAIN-701 Protocol Schedule Events (Protocol [Amendment 3] 24 October 2020) Table 2

| 1 | | SCR | SCR Cycle 1 (Day) | Cycle 1 (Day) | (Day) | | | Cycle 2 (Day) | (Day) | | Cycle 2 (Day) Cycles 3+ (Day | cles 3 | Cycles 3+ (Day) | ) (A | OBX | $EOT^1$ | FUP |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| X | Schedule of Events | | 1 | ∞ | 15 | 22 | | ∞ | 15 | | 1 | <b>∞</b> | 15 | 22 | | | |
| X | Informed Consent | × | | | | | | | | | | | | | | | |
| X | Eligibility | X | | | | | | | | | | | | | | | |
| X | Medical/Disease History/ | X | | | | | | | | | | | | | | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Smoking History | | | | | | | | | | | | | | | | |
| X | Demographics | X | | | | | | | | | | | | | | | |
| X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Physical Examination | X | × | | | | × | | | | × | | | | | × | X |
| X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | ECOG | X | × | | | | | | | | | | | | | | |
| tytusion X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X< | Weight | X | × | | | | × | | | | × | | | | | × | X |
| ead)³ X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X <th>Vital Signs</th> <th>X</th> <th></th> <th></th> <th></th> <th></th> <th></th> <th></th> <th></th> <th></th> <th></th> <th></th> <th></th> <th></th> <th></th> <th>×</th> <th>X</th> | Vital Signs | X | | | | | | | | | | | | | | × | X |
| EOI X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Pre-infusion | | × | × | × | × | × | × | × | × | × | × | × | × | | | |
| ead)³ X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X <td>EOI</td> <td></td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td></td> <td></td> <td></td> | EOI | | × | × | × | × | × | × | × | × | × | × | × | × | | | |
| ead) <sup>3</sup> X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X </th <td><math>30</math>, <math>60</math>, and <math>90</math> min after <math>EOI^2</math></td> <td></td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td>×</td> <td></td> <td></td> <td></td> | $30$ , $60$ , and $90$ min after $EOI^2$ | | × | × | × | × | × | × | × | × | × | × | × | × | | | |
| tylusion X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Electrocardiogram (12-lead) <sup>3</sup> | X | | | | | | | | | | | | | | × | X |
| FOI = X | Pre-infusion | | × | × | × | × | × | × | × | × | × | × | × | × | | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | EOI | | × | × | × | × | × | | | | | | | | | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | $I$ h after $EOI^2$ | | × | × | × | × | × | | | | | | | | | | |
| rededed² X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X< | $2 h after EOI^2$ | | × | × | × | × | × | × | × | × | × | × | × | × | | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | 3 h after EOf | | × | × | × | × | × | | | | | | | | | | |
| reeded <sup>2</sup> | $4 h after EOI^2$ | | × | × | × | × | × | × | × | × | × | × | × | × | | | |
| | hourly thereafter as needed <sup>2</sup> | | × | × | × | × | × | × | × | × | × | × | × | × | | | |
| | Hematology Panel | X | × | | | | × | | | | × | | | | | × | X |
| | Serum Chemistry Panel | X | X | X | X | × | X | × | × | × | X | × | X | X | | X | X |

<sup>&</sup>lt;sup>1</sup> Day 1 of Cycles 2+ and EOT Visit are Day 28 of the prior cycle
<sup>2</sup> For subjects with Grade 3 QTcF prolongation (≥ 501 msec or 60 msec increase compared to pre-infusion), repeat ECG every 15 to 30 minutes until resolved to Grade 2 (481 to 500 msec) or lower (≤ 499 msec) and then obtain ECGs every hour. If QTcF prolongation is ≥ Grade 3, an ECG may need to be repeated more frequently during a subject's visit as indicated in Table 6 , depending on the degree of the prolongation and per institutional standards.  $^3$  For subjects with  $\geq$  Grade 3 ( $\geq$  500 msec) QTcF prolongation with current or prior infusion

| 1 9 1 1 0 | SCR | ) | Cycle 1 (Day) | (Day) | | $\circ$ | Cycle 2 (Day) | (Day) | | Cy | cles 3- | Cycles 3+ (Day) | ( | OBX | $EOT^1$ | FUP |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Schedule of Events | | 1 | <b>∞</b> | 15 | 22 | 1 | <b>∞</b> | 15 | 22 | 1 | ∞ | 15 | 22 | | | |
| Serum Potassium | | | | | | | | | | | | | | | | |
| EOI | | × | | | | × | | | | | | | | | | |
| $3 h after EOI^2$ | | × | | | | × | | | | | | | | | | |
| Urinalysis | × | × | × | × | × | × | | | | × | | | | | | × |
| Pregnancy Test <sup>4</sup> | × | × | | | | × | | | | × | | | | | × | |
| PK Samples | | | | | | | | | | | | | | | | |
| Pre-infusion <sup>6</sup> | | × | | | | × | | | | | | | | | | |
| $EOI^6$ | | × | | | | × | | | | | | | | | | |
| 3 h after EOI <sup>6</sup> | | × | | | | × | | | | | | | | | | |
| 7 h after EOI <sup>6</sup> | | X <sub>7</sub> | | | | | | | | | | | | | | |
| at optional tumor biopsy | | | | | | | | | | | | | | X <sub>5</sub> | | |
| Biomarker Sample | | X | | | | X | | | | | | | | Χ <sub>2</sub> | X | |
| Potassium Supplementation <sup>8</sup> | | × | X | × | × | × | × | × | × | × | × | × | × | | | |
| Tarloxotinib Infusion | | × | × | × | × | × | × | × | × | × | × | × | × | | | |
| Tumor Tissue | × | | | | | | | | | | | | | | | |
| Optional Tumor Biopsy | | | | X5 | | | | | | | | | | X | X <sub>9</sub> | |
| Tumor Assessment | × | | Ţ | $\leftarrow$ Every 8 weeks (± 5 days) from Cycle 1 Day 1 $\rightarrow$ | ry 8 we | eks (± | 5 day | s) fron | Cycle | 1 Day | v 1 → | | | | | |
| Concomitant Medications | × | | | | | Ţ | ← Every Visit → | Visit – | <b></b> | | | | | × | × | |
| Adverse Events Assessment | | | | | | Ţ | $\leftarrow$ Every Visit $\rightarrow$ | Visit – | <b> </b> | | | | | × | × | × |

Abbreviations: CT = computed tomography; ECOG = Eastern Cooperative Oncology Group; EOI = end of infusion; EOT = End-of-Treatment Visit; FUP = Follow-up Visit; MRI = magnetic resonance imaging; OBX = optional biopsy; PET = positron emissions tomography; PK = pharmacokinetic; QTcF = corrected QT interval as calculated according to Fridericia's formula; SCR = Screening Period

 $<sup>^4</sup>$  Serum pregnancy at baseline, then urine dipstick, for women of childbearing potential.  $^5$  Collect blood (plasma samples for PK and biomarker including ctDNA) at time of biopsy  $^6$  Can be made  $\pm 5$  minutes of scheduled event.

<sup>&</sup>lt;sup>7</sup> In a subset of subjects.

<sup>&</sup>lt;sup>8</sup> If applicable, see Section 6.2.2.
<sup>9</sup> Collect blood (plasma sample for biomarker) at time of biopsy

#### 7 SAMPLE SIZE AND POWER

The primary objective of this study is to determine if tarloxotinib provides a clinically significant tumor response to subjects in each cohort, investigated by assessing if the true ORR is at least above some desirable target level following therapy with tarloxotinib.

According to the protocol, a Simon's 2-stage minimax design (Simon 1989) was used for all cohorts. The null hypothesis that the true response rate is 15% was tested against a one-sided alternative. In the first stage, 21 subjects were accrued. If there were 3 or fewer responses among these 21 subjects, the cohort was stopped for futility. Otherwise, 22 additional subjects may be accrued for a total of 43 subjects in each cohort. The null hypothesis will be rejected if 11 or more responses are observed in 43 subjects. This design yields a type I error rate of 0.0454 and power of 0.8014 when the true response rate is 31%. The probability of early termination at the end of the first stage is 0.61 if the true response rate is 15%.

#### 8 ANALYSIS SETS

## 8.1 Intent-To-Treat Analysis Set

The Intent-To-Treat (ITT) Analysis Set will include all enrolled subjects regardless of Treatment Period eligibility or completion. The ITT Analysis Set will be the basis for demographics and baseline characteristics. Since enrolled subjects are subjects who received at least one dose of tarloxotinib, the ITT Analysis Set is functionally the same as the Primary Analysis Set.

## 8.2 Primary Analysis Set

The Primary Analysis Set (PAS), referred to as the Safety Population in the protocol, is defined as all subjects who subjects who received at least 1 dose of tarloxotinib. The Primary Analysis Set will be the analysis population for the safety and efficacy analyses.

#### 9 GENERAL CONSIDERATIONS

#### 9.1 Presentation of Summary Statistics

For most summary statistics, data will be analyzed and displayed in tabular format. Continuous and categorical data will be summarized by cohort and overall.

Continuous variables will be summarized using a 6-point descriptive summary (n, mean, standard deviation [SD], median, minimum, and maximum) unless otherwise specified. The same number of decimal places as in the observed value will be presented when reporting minimum and maximum; 1 additional decimal place than in the observed value will be presented when reporting mean, median, 95% confidence interval (CI); 2 additional decimal places than in the observed value will be presented when reporting stable disease (SD).

All categorical/qualitative data will be presented using the frequency of events and percentages. All percentages will be presented to 1 decimal place, unless otherwise specified. Percentages equal to 100 will be presented as 100% and percentages will not be presented for zero frequencies. For summaries of AEs and CMs, the percentages will be based on the number of subjects who received study drug.

The statistical test for efficacy endpoints will not be performed.

Results of statistical analyses will be reported using summary tables, listings, and figures (TLFs). The ICH of Technical Requirements for Pharmaceuticals for Human Use numbering convention will be used for all TLFs.

All analyses and summaries will be produced using SAS® version 9.4 or higher.

#### 9.2 Definitions and Derived Variables

## 9.2.1 Screened and Enrolled Subjects

#### 9.2.1.1 Screened Subjects

Subjects who signed an informed consent form are considered Screened Subjects

## 9.2.1.2 Enrolled Subjects

Subjects who received at least one dose of tarloxotinib, are considered Enrolled Subjects.

## 9.2.2 Study Day

Study Day, which follows the CDISC Study Data Tabulation Model standard, is defined as (Assessment date - date of first study drug dosing + 1 day), where the assessment date is on or

after the date of first study drug dosing; (Assessment date - date of first study drug dosing), where the assessment date is before the date of first study drug dosing.

## 9.2.3 End of Study Treatment Definition

A subject is considered to have completed study treatment if the subject has completed the End of Treatment Visit.

## 9.2.4 End of Study Definition

A subject is considered to have completed the study if the subject has completed final safety follow-up visit. The end of the study is defined as the date of the last follow up visit of the last subject in the study.

#### 9.2.5 Date Last Known Alive

If a subject died, the date last known alive is the subject's date of death. Otherwise, the date last known alive is the date of last contact with the subject in the study (e.g., the most recent date of any in-clinic visit, date of telephone contact, date of withdrawal of consent, date of study completion date, etc.).

#### 9.2.6 Age

Age (years) will be calculated as the number of years between date of birth and date of the earliest informed consent, rounded down to the largest to a whole number less than or equal to the age at measurement.

#### 9.2.7 Body Mass Index

Body mass index  $(kg/m^2)$  is derived as weight (kg) / [height (m) × height (m)].

#### 9.2.8 Baseline Values

Baseline values are defined as the last, non-missing assessment prior to the first dose of study drug.

#### 9.2.9 Sum of Target Lesions

The sum of target lesions is defined as the sum of the longest diameters for non-nodal lesions and the short axis for lymph nodes.

## 9.2.10 Evaluable Subjects

A subject is classified as response evaluable if they have at least one response assessment or if they discontinue from treatment due to death prior to obtaining at least one response assessment. Subjects discontinuing treatment for disease progression must have a disease assessment performed documenting the progression

## **9.2.10.1 Responder**

All enrolled subjects who receive study treatment, have a baseline tumor assessment with documentation of measurable disease, have at least 1 on-study tumor assessment, whether or not this occurs at the specified imaging interval, will be considered evaluable for response. Subjects will be considered responders if they have a confirmed objective response of CR or PR according to RECIST v1.1 recorded from baseline until disease progression or death due to any cause.

## 9.2.11 RECIST Response Assessment

 Table 3
 Response Evaluation Criteria in Solid Tumours Guidelines

| Response assessment | RECIST guideline, version 1.1 |
|---|---|
| Target lesions | |
| Complete Response | Disappearance of all target lesions and reduction in the short axis measurement of all pathologic lymph nodes to $\leq$ 10 mm |
| Partial Response | ≥30% decrease in the sum of the longest diameter of the target lesions compared with baseline |
| Progressive Disease | ≥20% increase of at least 5 mm in the sum of the longest diameter of the target lesions compared with the smallest sum of the longest diameter recorded <b>OR</b> The appearance of new lesions, including those detected by fludeoxyglucose PET |
| Stable Disease | Neither partial response nor progressive disease |
| Non-target lesions | |
| Complete Response | Disappearance of all non-target lesions and normalization of tumor marker levels |
| Incomplete Response;<br>Stable Disease | Persistence of 1 or more non-target lesions and/or the maintenance of tumor marker levels above normal limits |
| Progressive Disease | The appearance of 1 or more new lesions or unequivocal progression |
| If subject has measurable disease, an increase in the overall level or sub-<br>worsening in non-target lesions, such that tumor burden has increased,<br>there is stable disease or partial response in target lesions | |

If no measurable disease, an increase in the overall tumor burden comparable in magnitude with the increase that would be required to declare progressive disease in measurable disease (eg, an increase in pleural effusions from trace to large, or an increase in lymphangitic disease from localized to widespread)

#### 9.2.11.1 Overall Response Rate

The overall response rate in each cohort will be estimated as the number of subjects with a confirmed objective response (CR or PR) divided by the number of enrolled subjects (defined in Section 9.2.10) in each respective cohort.

## 9.2.11.2 Best Overall Response Rate

Best overall response rate is calculated the same as the ORR (Section 9.2.11.1), but subjects are summarized at their best response level. Best to worst response is as follows: CR, PR, SD, and then PD.

## 9.2.12 Duration of Response

DOR as measured from the date of first objective response (CR or PR) to date of disease progression or death is documented. DOR data will be censored according to Table 4 for subjects who are alive with no objective documentation of (radiographic) disease progression by the data cut-date.

Table 4 Censoring Rules for Progression-Free Survival

| ole 4 Censoring Rules for 11 ogression-1 | i ce Sui vivai |
|---|---|
| Situation | Date of Censoring |
| No baseline radiologic assessment | Date of first study drug dose |
| No post-baseline radiologic assessment (and<br>no death prior to first scheduled radiologic<br>assessment) | Date of first study drug dose. |
| No progression or death on study | Date of last radiologic assessment |
| Documented progression or death after 2 or more consecutive missing radiologic assessments | Date of last radiologic assessment |
| New anticancer therapy started prior to | Date of last radiologic assessment prior to |
| progression | new anticancer therapy |

#### 9.2.13 Disease Control Rate

Disease control rate is defined as the number of subjects who have CR, PR, or SD for at least 2 cycles (8 weeks) according to the RECIST v1.1 recorded in the period between first study drug dose and disease progression or death to any cause. The DCR on each cohort will be estimated

by dividing the number of subjects with CR, PR, or SD for at least 2 cycles (8 weeks) by the number of subjects enrolled in each cohort.

## 9.2.14 Progression-Free Survival

Progression-free survival is defined as the time from the date of first tarloxotinib dose to the date of the first objective documentation of radiographic disease progression or death due to any cause, whichever occurs first. PFS data will be censored according to Table 4 for subjects who are alive with no objective documentation of (radiographic) disease progression by the data cut-date.

#### 9.2.15 Overall Survival

Overall survival as measured from the date of first tarloxotinib dose to the date of death by any cause. In the absence of confirmation of death, survival time will be censored to last date the subject is known to be alive.

## 9.2.16 Study Drug Exposure Variables

## 9.2.16.1 Total Tarloxotinib Dose (mg) Taken

Total tarloxotinib dosage (mg) is defined as the cumulative dosage of tarloxotinib actually received over the Treatment Period, calculated as follows:

$$Total\ Tarloxotinib\ Dose = \sum_{i=1}^{k} (Actual\ Tarloxotinib\ Dose)_{i}$$

where

 $\Sigma$  represents the summation operator and the value in parentheses is summed over the sequence i = 1 to k, where k = number of tarloxotinib infusions subject received.

## 9.2.16.2 Actual Number of Infusions Administered

The number of infusions a subject received. Interrupted infusions also count as one infusion.

## 9.2.16.3 Actual Number of Cycles Administered

The number of cycles a subject initiated. This includes receiving infusions at each scheduled visit of the cycle (Day 1, Day 8, Day 15, and Day 22).

## 9.2.16.4 Actual Dose Intensity

Actual dose intensity (mg/day) is calculated as total cumulative dose received divided by actual number of infusions administered.

#### 9.2.16.5 Treatment Duration

Treatment duration (days) is defined as (Last Dose Date – First Dose Date + 1 day). Treatment duration indexed by the 28-day cycles is defined as ([Last Dose Date – First Dose Date + 1 day]/28 days), rounded to one decimal place.

## 9.2.17 Prior, Concomitant and Post treatment Medications

All medication verbatim terms reported on the electronic case report form (eCRFs) will be mapped according to the World Health Organization (WHO) Drug Dictionary (WHO DD March 2020 B3). The medications will be mapped to Anatomical/Therapeutic/Chemical (ATC) class and preferred names.

A prior medication is considered to be any medication that is taken within a year prior to the first study drug dosing.

A concomitant medication is considered to be any medication that is continued from Screening and continued after the first study drug dosing (i.e., a prior medication can also be a CM if it continued after the first dose of study drug) or any medication with start dates or stop dates within the Treatment Period. Specifically, CMs are medications: that are continued from Screening and continued after the first study drug dosing, or with start dates or stop dates within the first dose date through last dose date + 24 hours, missing CM end date, or ongoing) with the study drug administration.

Post medications is considered to be any medication taken after the last study drug dose date + 24 hours, missing CM end date, or ongoing.

#### 9.2.18 Adverse Events

All AE verbatim terms reported on the eCRFs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA® version 22.0). AE severity will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE

2017) version 5. MedDRA will be used to map the AE verbatim to lowest level term, preferred term, and system organ class for summary purposes.

 Table 5
 Severity Grading Guideline for Adverse Events

| Grade | Description |
|-------|----------------------------------------------------------|
| 1 | Mild; Asymptomatic or mild symptoms; Clinical or |
| | diagnostic observations only; Intervention not indicated |
| 2 | Moderate; Minimal, local or noninvasive intervention |
| | indicated; Limiting age-appropriate instrumental |
| | activities of daily living* |
| 3 | Severe or medically significant but not immediately |
| | life-threatening; Hospitalization or prolongation of |
| | hospitalization indicated; Disabling; Limiting self-care |
| | activities of daily living <sup>†</sup> |
| 4 | Life-threatening consequences; Urgent intervention |
| | indicated |
| 5 | Death related to adverse event |

## 9.2.18.1 Treatment-Emergent Adverse Events

Treatment-emergent adverse events are defined as any AEs, regardless of relationship to study drug, that have an onset or worsening in severity on or after the first dose of study drug until 30 days after the final dose of study drug (safety follow-up visit).

Related TEAEs are those reported by investigators as related to the study drug.

## 9.2.18.2 Serious Adverse Events

Serious AEs are defined according to the NCI CTCAE v5.0, as described in Protocol Section 8.2.2 Adverse Event Severity.

#### 9.2.18.3 Severe Adverse Events

Severe AEs are defined as events with a severity of Grade 3 or higher.

\* Instrumental activities of daily living refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

<sup>†</sup> Self-care activities of daily living refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden

## 9.2.18.4 Serious Unexpected Suspected Adverse Reaction

A serious AE deemed related to the study drug (adverse reaction) is considered "unexpected" if it is not listed in the Investigator's Brochure (i.e., ECG QT prolonged, Hypertension, Rash [rash, infusion site rash and rash erythematous]) or is not listed at the specificity or severity that has been observed.

#### 9.3 Analysis Windows

Clinical visits may occur outside protocol-specified windows. Therefore, instead of relying solely on visit labels in the clinical database, analysis visits and their windows are defined using Study Day (See Section 9.2.2). For the purposes of data analysis and summary, assessments and/or measurements will be flagged based on the collection date/time that is closest to the protocol-scheduled time point (or target Study Day). Analysis visit windows are presented in by type of assessments and/or measurements.

**Table 6** Visit Analysis Windows (Clinic visits only)

| Protocol<br>Specified Visit | Target Study Day | Start (days) | Stop (days) |
|-----------------------------|------------------|--------------|-------------|
| Screening | -114 | low | -1 |
| Cycle 1 Day 1 | 1 | 1 | 4 |
| Cycle 1 Day 8 | 8 | 5 | 11 |
| Cycle 1 Day 15 | 15 | 12 | 18 |
| Cycle 1 Day 22 | 22 | 19 | 25 |
| Cycle 2 Day 1 | 29 | 26 | 32 |
| Cycle 2 Day 8 | 36 | 33 | 39 |
| Cycle 2 Day 15 | 43 | 40 | 46 |
| Cycle 2 Day 22 | 50 | 47 | 53 |
| Cycle 3 Day 1 | 57 | 54 | 60 |
| Cycle 3 Day 8 | 64 | 61 | 67 |
| Cycle 3 Day 15 | 71 | 68 | 74 |
| Cycle 3 Day 22 | 78 | 75 | 81 |
| Cycle 4 Day 1 | 85 | 82 | 88 |
| Cycle 4 Day 8 | 92 | 89 | 95 |
| Cycle 4 Day 15 | 99 | 96 | 102 |
| Cycle 4 Day 22 | 106 | 103 | 109 |
| Cycle 5 Day 1 | 113 | 110 | 116 |
| Cycle 5 Day 8 | 120 | 117 | 123 |
| Cycle 5 Day 15 | 127 | 124 | 130 |
| Cycle 5 Day 22 | 134 | 131 | 137 |

| Protocol<br>Specified Visit | Target Study Day | Start (days) | Stop (days) |
|---|---|---|---|
| Cycle 6 Day 1 | 141 | 138 | 144 |
| Cycle 6 Day 8 | 148 | 145 | 151 |
| Cycle 6 Day 15 | 155 | 152 | 158 |
| Cycle 6 Day 22 | 162 | 159 | 165 |
| Cycle 7 Day 1 | 169 | 166 | 172 |
| Cycle 7 Day 8 | 176 | 173 | 179 |
| Cycle 7 Day 15 | 183 | 180 | 186 |
| Cycle 7 Day 22 | 190 | 187 | 193 |
| Cycle 8 Day 1 | 197 | 194 | 200 |
| Cycle 8 Day 8 | 204 | 201 | 207 |
| Cycle 8 Day 15 | 211 | 208 | 214 |
| Cycle 8 Day 22 | 218 | 215 | 221 |
| Cycle 9 Day 1 | 225 | 222 | 228 |
| Cycle 9 Day 8 | 232 | 229 | 235 |
| Cycle 9 Day 15 | 239 | 236 | 242 |
| Cycle 9 Day 22 | 246 | 243 | 249 |
| Cycle 10 Day 1 | 253 | 250 | 256 |
| Cycle 10 Day 8 | 260 | 257 | 263 |
| Cycle 10 Day 15 | 267 | 264 | 270 |
| Cycle 10 Day 22 | 274 | 271 | 277 |
| End of Treatment | Treatment End<br>Date | Study Day <=<br>(ADSL.TRTEDT -<br>ADSL.TRTSDT + 1) | |
| Follow-up | Treatment End<br>Date + 30 Days (± 7<br>days) | Study Day ><br>(ADSL.TRTEDT -<br>ADSL.TRTSDT + 1) | high |

## 10 STATISTICAL AND ANALYSIS ISSUES

## **10.1** Adjustments for Covariates

No adjustments for covariates will be performed in the study.

## 10.2 Handling Dropouts or Missing Data

Missing data will not be imputed. Every effort will be made by the Sponsor to ensure completeness of data collection.

## 10.2.1 Handling of Laboratory Data

A retest value will be used if the first test is invalidated, e.g., specimen hemolyzed.

## 10.2.2 Handling of Safety Data

#### 10.2.2.1 Adverse Events

If the time of onset (before or after intake of study drug) cannot be determined whether an AE is treatment-emergent because of a partial onset date, the event will be counted as a TEAE.

Adverse events with incomplete start dates will be considered TEAEs, if:

- Day and month are missing and the year is equal to or after the year of the first date of study drug dosing;
- Month is missing and the year is after the year of the first date of study drug dosing;
- Day is missing and the year is equal to the year of the first date of study drug dosing and the month is equal to or after the month of the first date of study drug dosing; or
- Year is missing.

If severity or relationship of an AE to study drug is not recorded, the severity or relationship will be imputed as "severe" or relationship as "possibly related," for analysis purposes.

#### 10.2.2.2 Concomitant Medications

If start date of a medication is missing, the medication will be considered to have started prior to the study. Such a medication may also be considered concomitant, depending on the stop date or lack thereof. If the stop date of a concomitant medication is missing, then the medication will be treated as ongoing. If the start date of a medication is missing, the stop date will be used to determine whether or not it is concomitant. Medications with other incomplete start dates or end dates will be imputed as follows:

Incomplete medication start date/time:

- If only have a YEAR, impute as Jan. 1.
- Else if only have YEAR and MONTH, impute as Day 1 of month.
- Otherwise missing, no imputation.

Incomplete medication end date/time:

- If only have a YEAR, impute as December 31.
- Else if only have YEAR and MONTH, then impute to last day of the month.
- Otherwise missing, no imputation.

## 10.3 Multicenter Considerations

This trial will be conducted at 14 study centers in the United States, Canada, and other regions. Data from all study centers will be pooled for efficacy and safety analyses. Because the number of subjects at each center is likely to be small, no analyses will be performed by center. Subjects from all centers will be pooled for all analyses.

#### 10.4 Multiple Comparisons, Multiplicity

Efficacy variables will be assessed without adjustment for multiple comparisons.

#### 10.5 Active-Control Studies

There is no comparator in this study as all subjects are treated with tarloxotinib.

## 10.6 Examination of Subgroups

Efficacy variables will be assessed without examination of subgroups.

#### 11 STUDY SUBJECTS

#### 11.1 Subject Enrollment and Disposition

#### 11.1.1 Enrolled Subjects

An accounting of the study subjects will be tabulated. Subjects not completing the study will be listed along with the reason for their premature discontinuation. Reasons for premature discontinuation will be summarized.

Enrolled (Section 9.2.1) subjects will be summarized by cohort and overall.

#### **Treatment Periods**

- Number of subjects enrolled (ITT)
  - o Number (%) of subjects who discontinued from the study treatment
    - The primary reason for withdrawal from the study treatment
  - o Number (%) of subjects who completed the study
  - O Number (%) of subjects who discontinued from the study
    - ➤ The primary reason for withdrawal from the study

The percentages will be based on the total subjects who are enrolled (ITT).

A listing of disposition will be provided for all enrolled subjects.

#### 11.2 Protocol Deviations

Protocol deviations will be neither listed nor summarized because RAIN-701 was discontinued and this SAP will support an abbreviated clinical study report, which does not include protocol deviations per FDA guidance (Food and Drug Administration, 1999).

## 11.3 Demographics and Baseline Characteristics

Demographics and baseline characteristics will be summarized and listed for all treated subjects (ITT). Demographic characteristics will include age, sex, race, and ethnicity. A subject listing of demographics will be provided.

## 11.3.1 Key Baseline Demographics

The following parameters from each of the individual baseline and historical summaries will be summarized in a single summary:

- Age
- Age group, n (%)
- Sex, n (%)
- Race, n (%)
- Ethnicity, n (%)
- Smoking status, n (%)
- Baseline weight (kg)
- ECOG performance status, n(%)
- Mutation status, n (%)
- Stage at time of disease, n (%)
- Stage at time of study entry, n (%)

#### 11.4 Medical History

Medical history and current medical conditions will be mapped to preferred terms and system organ classes using the MedDRA® Dictionary (version 23.0) Medical history will be summarized by system organ class (SOC) and preferred term (PT) by cohort and overall for ITT subjects. A subject listing of general medical history will include start date/end date, verbatim medical history term, SOC, PT, and ongoing status (Yes, No). Additional subject listings of prior radiation therapy and prior surgeries will contain the start date and end date (if available) and

type of procedure. The subject listing of prior systemic therapies will include at a start date, end date, medication, reason the therapy ended, and best overall response.

#### 12 STUDY DRUG AND OTHER MEDICATIONS

#### 12.1 Exposure to Study Drug and Study Treatment Compliance

Summaries of study drug exposure and compliance will be summarized overall and by cohort. The source for study drug dosing and compliance is drug exposure.

The summaries will include total number of cycles initiated, the median (range) of cycles administered, and dose intensity (see definitions in Section 9.2.11) by cohort and overall. The denominators for percentages will be the number of subjects who received the study treatment.

#### 12.2 Prior and Concomitant Medications

Prior and concomitant medications (see definition in Section 9.2.10), will be summarized using WHO DD ATC class and preferred name. The summary results will be presented by cohort. Prior medications will be summarized by cohort. Concomitant medications will be summarized by cohort and overall.

These summaries will present the number and percentage of subjects using each medication. Subjects may have more than one medication within an ATC class and preferred name. At each summary level subjects are counted once if they reported one or more medications at that level. Each summary will be ordered by descending frequency of incidence of ATC class and preferred name within each ATC class.

All medications will be provided in a subject listing with flags indicating study drug dose level. The variables include, but not limited to: Start date/end date/ongoing, medication name, ATC class and preferred name, indication, dose, unit, form, frequency, and route.

#### 13 EFFICACY ANALYSES

## 13.1 Primary Analysis

The primary analysis was planned after all subjects stop tarloxotinib treatment until documented disease progression or unacceptable toxicity. The primary analysis will not be performed because RAIN-701 was discontinued and this SAP supports an abbreviated clinical study report. Additionally, efficacy analyses are unlikely to be significant because the sample size is small and the analyses will be underpowered. In place of formal primary analyses, selected efficacy endpoints will be summarized descriptively.

## 13.2 Primary Efficacy

The primary objective of this study is to evaluate the ORR of tarloxotinib as defined as a CR or PR according to RECIST v1.1 recorded from baseline until disease progression or death due to any cause.

The numbers and percentages of subjects meeting each response will be summarized, and the ORR will be summarized by cohort along with the corresponding 2-sided 95% CI calculated using the binomial exact method. All treatment responses and all tumor assessments will be listed.

The maximum percent reduction from baseline in the sum of target lesions will be displayed as a waterfall plot. The waterfall plot will have a y-axis that will be the maximum percent change from baseline in the sum of target lesions, and the x-axis will be each cohort and overall.

The best overall response (Section 13.3) will be reported similarly.

#### 13.3 Secondary Efficacy

The secondary efficacy objective is to evaluate further measures of antitumor activity of tarloxotinib including:

- Best overall response (Reporting as described in Section 13.2),
- Duration of response (Section 13.3.1),
- Disease control rate (Section 13.2),

- Progression-free survival (Section 13.3.2), and
- Overall survival (Section 13.3.2)

The additional secondary objectives of exploratory biomarkers of hypoxia in tumor tissue and plasma exposure to tarloxotinib and effects on cardiac repolarization will not have analyses or descriptive summarization of these endpoints due to the limited data basis.

#### 13.3.1 Duration of Response

DOR will be summarized using descriptive statistics (Section 9.1) for each cohort and overall. The DOR data will be listed for each subject.

#### 13.3.2 Survival Reporting

The PFS and OS will be summarized using the Kaplan-Meier method and displayed graphically by cohort and overall: Median event times and the corresponding 2-sided 95% CI will be provided. The number and % of subjects with disease progression or death will be provided. The number and % of subjects censored as well as reasons for censoring will be provided. A listing of survival data will be provided.

#### 13.4 Exploratory Objectives

The exploratory objectives are:

- To evaluate the concordance of EGFR mutation, HER2 mutation, and NRG1, EGFR,
   HER2, and HER4 fusion detection between tissue and plasma using ctDNA
- To evaluate exploratory biomarkers of hypoxia in tumor tissue including 6
   transmembrane epithelial antigen of the STEAP4 expression and ERBB family and cancer cell signaling pharmacodynamic markers
- To evaluate the pharmacokinetics of tarloxotinib and tarloxotinib-E in tumor tissue

Analysis and descriptive summary of these exploratory endpoints are outside the scope of this SAP.

#### 13.5 Subgroup Analyses

No examination of subgroups is planned.

#### 14 SAFETY ANALYSES

One of the study objectives is to assess the safety of tarloxotinib. Safety will be assessed by repeated clinical evaluations including adverse events (AEs), serious AEs (SAEs), suspected serious unexpected suspected adverse reactions, vital signs, physical examination, electrocardiograms (ECGs), clinical laboratory tests (serum chemistry, hematology, and urinalysis). All analyses of the safety data will be performed using the primary analysis set. All descriptive statistics (described in Section 9.1) will be presented by cohort and overall.

#### 14.1 Adverse Events

Safety will be assessed by repeated clinical evaluations including adverse events (AEs), serious AEs (SAEs), serious unexpected suspected adverse reactions (SUSARs), and deaths.

Safety data will be summarized descriptively. AEs will be summarized by severity, seriousness, and relationship to study drug. All AEs including the AE verbatim term and the associated AE MedDRA preferred term will be provided in the subject data listings. Incidence of treatment-emergent AEs will be summarized descriptively by cohort and total.

TEAEs are defined in Section 9.2.18.1. All reported AEs (including non-TEAEs) will be listed. Separate listings will be provided for suspected adverse reactions, unexpected events, SAEs, and serious unexpected suspected adverse reactions. All TEAE summary tables will present the number and percentages of subjects reporting TEAEs, unless otherwise specified. A summaries of TEAEs by severity, seriousness, and relation to study drug will be tabulated.

## 14.1.1 Overall Summary of TEAEs

Overall summary of TEAEs will be presented by cohort and overall. Subjects will be counted only once at the highest severity when summarizing TEAE by severity. The overall summary will include the following:

- Number (%) of subjects with any TEAEs
- Number (%) of subjects with any TEAEs by severity
- Number (%) of subjects with any serious TEAEs
- Number (%) of subjects with any related TEAEs
- Number (%) of subjects with any serious unexpected suspected adverse reactions
- Number (%) of subjects with any TEAEs leading to study drug discontinuation
- Number (%) of subjects with any AEs leading to death

#### 14.1.2 Summary of TEAEs by System Organ Class and Preferred Term

AEs will be summarized by MedDRA SOC and PT. Subjects can experience more than one AE per SOC and PT. At each level of subject summarization (SOC or PT or severity), subjects will be counted once if they reported at least one AE at that level (SOC or PT or severity). Each summary will be ordered by SOC alphabetically and by PT in descending order of the total incidence within each SOC. Summary tables will be created for each of the following types of AEs:

- TEAEs
- Severe (≥ Grade 3) TEAEs
- Related TEAEs
- TEAEs leading to study drug discontinuation
- Serious TEAEs
- Serious unexpected suspected adverse reactions
- TEAEs leading to death

#### 14.1.3 Summary of TEAEs by Preferred Term

AEs will be summarized by MedDRA preferred term (PT). Subjects can experience more than one AE per PT. At each preferred term, subjects will be counted once if they reported at least one AE at that level (PT). Each summary will be ordered by PT in descending order of the incidence. Summary tables will be created for each of the following types of AEs:

- TEAEs
- Severe (≥ Grade 3) TEAEs
- Related TEAEs
- TEAEs leading to study drug discontinuation
- Serious TEAEs
- Serious unexpected suspected adverse reactions
- TEAEs leading to death

#### 14.2 Clinical Laboratory Evaluation

Results for clinical laboratory parameters (serum chemistry and hematology), vital signs, ECGs, and physical examinations will be summarized by cohort and combined and by study visits.

Descriptive summary statistics in observed values as well as changes from baseline will be

presented. In addition, thresholds of marked laboratory abnormalities based on NCI CTCAE v5.0 will be summarized by worst grade shift from baseline (see Appendix B).

Table 7 shows clinical laboratory assessments (hematology, chemistry, and urinalysis) that were performed performed. Chemistry and hematology laboratory parameters will be summarized by cohort and scheduled visit. Urinalysis assessments will be listed but not summarized due to their qualitative nature.

**Table 7** Clinical Laboratory Parameters

| Chem | istry | Hematology | Urinalysis |
|---|---|---|---|
| Sodium | Creatinine | Hematocrit | Specific gravity |
| Potassium | Total Bilirubin | Hemoglobin | Protein |
| Chloride | AST/SGOT | WBC count | Glucose |
| Bicarbonate | ALT/SGPT | Neutrophils | Ketones |
| Calcium | <del>ALP</del> ‡ | Lymphocytes | Urobilinogen |
| Magnesium | Albumin | Monocytes | Occult blood |
| Phosphorous | Total protein | Eosinophils | Microscopic sediment |
| | | | evaluation <sup>‡</sup> |
| Glucose | | Basophils | |
| Blood urea nitrogen | | Platelet count | WOCBP only: |
| | | | β-HCG§ |

ALT = alanine aminotransferase; ALP = alkaline phosphatase; AST = aspartate aminotransferase; HCG = β-human chorionic gonadotropin pregnancy; SGOT = serum glutamic-oxaloacetic transaminase; SGPT = serum glutamic pyruvic transaminase; WBC = white blood count; WOCBP = women of child-bearing potential

Numeric results will be summarized using (6-point) descriptive statistics at baseline and at each scheduled post-baseline time point, unless otherwise specified. Changes from baseline will also be summarized by scheduled time point, where available. Selected laboratory results will be listed with CTCAE reference ranges.

#### 14.3 Vital Signs

Descriptive statistics for pulse rate, respiratory rate, temperature, weight, and blood pressure (systolic and diastolic) including baseline values and change from baseline values, will be summarized by cohort and scheduled time point. All vital signs parameters will be listed.

<sup>‡</sup> Alkaline phosphatase and microscopic sediment evaluation will neither be listed nor summarized due to lack of data § β-HCG pregnancy test may be collected as a serum, urine, or urine dipstick assessment

#### 14.4 12-Lead Electrocardiogram

Electrocardiogram (ECG) data, such as clinical interpretation of ECGs, heart rate (HR) values, and interval assessments of QRS duration, PR interval, QT interval, and the Fridericia's corrected value of the interval between the Q and T waves on the ECG tracing (QTcF) will be listed. Descriptive statistics for observed values and change from baseline at each scheduled time point will be presented for these 12-lead ECG interval and HR assessments will be presented as actual values and as changes from the baseline values by 6-point descriptive summary statistics (n, mean, SD, median, minimum, and maximum). The numbers and percentages of subjects who meet categorical analyses such as the following criteria at each scheduled ECG time point will be presented.

- Absolute QTcF interval:
  - o QTcF interval < 450
  - o QTcF interval 451 to 480 msec
  - o QTcF interval 481 to 500 msec
  - o QTcF interval  $\geq$  501 msec
- Change from predose baseline in QTcF interval:
  - $\circ \le 30 \text{ msec}$
  - o 31 to 60 msec
  - o 60 msec

The numbers and percentages of subjects meeting each criterion will be summarized for each ECG time point, as well as for each subject overall at any time.

Abnormal ECG findings not present at the pre-dose baseline will be summarized as the number of subjects with each finding at 1 or more ECG times. Descriptive waveform morphology changes will be provided.

#### 15 CHANGES RELATIVE TO THE PROTOCOL-SPECIFIED ANALYSIS

Protocol Section 9.2.3 states "Deviations will be defined prior to database lock. Handling of major deviations in statistical analyses will be defined in the SAP" and further defines a Per-Protocol analysis set excludes subjects with certain, pre-specified deviations. RAIN-701 was terminated and the analysis will support an abbreviated clinical study report, which does not include protocol deviations per FDA guidance for industry, Submission of Abbreviated Reports and Synopses in Support of Marketing Applications. Analysis will be performed on the safety population which includes all subjects who received at least 1 dose of tarloxotinib. Analysis of a Per Protocol (PP) population where subjects with major protocol deviations are removed is not necessary for the aCSR. The abbreviated CSR will provide a comprehensive safety analysis for all subjects receiving at least 1 dose of tarloxotinib. Additionally, the primary efficacy analysis of ORR will include all treated subjects. Efficacy analyses are not interpretable as RAIN-701 was terminated and did not enroll the intended sample size to support statistical analyses.

Protocol Section 7 states, "In accordance with RECIST v1.1, response (PR and CR) must be confirmed by a second tumor assessment at least 8 weeks after the initial observed response." SAP Section 6.3.1 text instead states that the confirmation assessment must be at least 4 weeks after the initial observed response, which is aligned with the true RECIST v1.1 criteria. The efficacy endpoint (Section 9.2.13) still follows the protocol text in defining the disease control for at least 8 weeks (2 cycles).

Protocol Table 12 states "Microscopic sediment evaluation, as clinically indicated" as a urinalysis assessment, but these microscopic sediment urinalysis assessments were not collected. Similarly, Protocol Table 12 lists ALP as a serum chemistry assessment, but it was not collected.

Units and reference ranges of the local laboratory assessments were not collected. The Sponsor has assigned units and lab normal ranges for each parameter (e.g., lower limit of normal, upper limit of normal) based on available information and Harrison's Principles of Internal Medicine (Appendix A).

Rain Therapeutics Inc. RAIN-701 SAP


Adverse events were coded with MedDRA version 22.0 and medical history events were coded with MedDRA version 23.0.

#### 16 References

- Cancer Therapy Evaluation Program. (2017, November 27). Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. National Institutes of Health National Cancer Institute, U.S. Department of Health and Human Services. Retrieved from CTEP: https://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/CTCAE\_v5\_Q uick\_Reference\_8.5x11.pdf
- Food and Drug Administration. (1999, September 13). Submission of Abbreviated Reports and Synopses in Support of Marketing Applications. Centers for Drug Evaluation and Research (CDER) and Biologics Evaluation and Research (CBER), U.S. Department of Health and Human Services. Rockville, MD: Federal Register. doi:99-23663
- International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use. (1996, July). *Structure and Content of Clinical Study Reports (ICH E3)*. Center for Drug Evaluation and Research (CDER), U.S. Department of Health and Human Services. Rockville, MD: Federal Register. doi:96-18000
- International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use. (1998, September). *Statistical Principles for Clinical Trials (ICH E9)*. Centers for Drug Evaluation and Research (CDER) and Biologics Evaluation and Research (CBER), U.S. Department of Health and Human Services. Rockville, MD: Federal Register. doi:98-24754

### 17 Appendix A: Local Laboratory Units and Reference Ranges by Site and Parameter When a reference range is followed by an asterisk, it is sourced from Harrison's Principles of Internal Medicine, 19<sup>th</sup> edition.

 Table 8
 Site 101 Units and Reference Ranges by Parameter

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 101 | Chemistry | Albumin | | | g/dL | 3.5 | 5 |
| 101 | Chemistry | ALP | | | /L | 45 | 117 |
| 101 | Chemistry | ALT/SGPT | | | /L | 15 | 41 |
| 101 | Chemistry | AST/SGOT | | | /L | 3 | 34 |
| 101 | Chemistry | Bicarbonate | | | mmol/L | 18 | 23 |
| 101 | Chemistry | Blood urea nitrogen | M | | mg/dL | 9 | 20 |
| 101 | Chemistry | Blood urea nitrogen | F | | mg/dL | 7 | 17 |
| 101 | Chemistry | Calcium | | | mmol/L | 1.12 | 1.32 |
| 101 | Chemistry | Chloride | | | mmol/L | 98 | 107 |
| 101 | Chemistry | Creatinine | M | | mg/dL | 0.66 | 1.5 |
| 101 | Chemistry | Creatinine | F | | mg/dL | 0.52 | 1.04 |
| 101 | Chemistry | Glucose | | | mg/dL | 65 | 140 |
| 101 | Chemistry | Magnesium | | | mg/dL | 1.6 | 2.3 |
| 101 | Chemistry | Phosphorous | | | mg/dL | 2.5 | 4.5 |
| 101 | Chemistry | Potassium | | | mmol/L | 3.5 | 5.1 |
| 101 | Chemistry | Sodium | | | mmol/L | 137 | 145 |
| 101 | Chemistry | Total Bilirubin | | | mg/dL | 0.2 | 1.3 |
| 101 | Chemistry | Total protein | | | g/dL | 6.3 | 8.2 |
| 101 | Hematology | Basophils | | | k/uL | 0 | 0.2 |
| 101 | Hematology | Eosinophils | | | k/uL | 0 | 0.7 |
| 101 | Hematology | Hematocrit | M | | % | 37.5 | 49.5 |
| 101 | Hematology | Hematocrit | F | | % | 34.5 | 44 |
| 101 | Hematology | Hemoglobin | M | | g/dL | 12.5 | 16.5 |
| 101 | Hematology | Hemoglobin | F | | g/dL | 11 | 14.5 |
| 101 | Hematology | Lymphocytes | | | k/uL | 0.6 | 4.9 |
| 101 | Hematology | Monocytes | | | k/uL | 0.1 | 1.3 |
| 101 | Hematology | Neutrophils | | | k/uL | 1.7 | 8.1 |
| 101 | Hematology | Platelet count | | | k/uL | 145 | 400 |

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 101 | Hematology | WBC count | | | k/uL | 4 | 10.8 |
| 101 | Urinalysis | Glucose | | | | Normal | |
| 101 | Urinalysis | Ketones | | | | Negative | |
| 101 | Urinalysis | Occult blood | | | | Negative | |
| 101 | Urinalysis | Protein | | | | Negative | |
| 101 | Urinalysis | Specific gravity | | | | 1.003 | 1.03 |
| 101 | Urinalysis | Urobilinogen | | | mg/dL | < 2.0 | |
| Table 9 | Site 102 Uni | ts and Reference | Range | s by P | arameter | | |
| SITE | | | C | | | REFERENCE | REFERENCE |
| NUMBER<br>102 | PANEL | PARAMETER Albumin | SEX | K AGI | | LOW 3.5* | HIGH 5.5* |
| | Chemistry Chemistry | ALP | | | g/dL | 3.3 | 3.3 |
| 102 | | | | | T T /T | 7* | 41* |
| 102 | Chemistry | ALT/SGPT<br>AST/SGOT | | | U/L | | |
| 102 | Chemistry | AS1/SGO1 Bicarbonate | | | U/L | 12* | 38* |
| 102 | Chemistry | | | | meq/L | 22*<br>7* | 30* |
| 102 | Chemistry | Blood urea nitrogen | | | mg/dL | · | 20* |
| 102 | Chemistry | Calcium | | | mg/dL | 8.7* | 10.2* |
| 102 | Chemistry | Chloride | Г | | meq/L | 102* | 109* |
| 102 | Chemistry | Creatinine | F | | mg/dL | 0.5* | 0.9* |
| 102 | Chemistry | Creatinine | M | | mg/dL | 0.6* | 1.2* |
| 102 | Chemistry | Glucose | | | mg/dL | 65* | 95* |
| 102 | Chemistry | Magnesium | | | mg/dL | 1.5* | 2.3* |
| 102 | Chemistry | Phosphorous | | | mg/dL | 2.7 | 4.5 |
| 102 | Chemistry | Potassium | | | meq/L | 3.5* | 5* |
| 102 | Chemistry | Sodium | | | meq/L | 136* | 146* |
| 102 | Chemistry | Total Bilirubin | | | mg/dL | 0.1 | 1.3 |
| 102 | Chemistry | Total protein | | | g/dL | 6.7* | 8.6* |
| 102 | Hematology | Basophils | | | 10^9/L | 0 | 0.2 |
| 102 | Hematology | Eosinophils | | | 10^9/L | 0 | 0.4 |
| 102 | Hematology | Hematocrit | M | | % | 39.2 | 50.2 |
| 102 | Hematology | Hematocrit | F | | % | 35.7 | 46.7 |
| 102 | Hematology | Hemoglobin | M | | g/dL | 14.3 | 18.1 |
| 102 | Hematology | Hemoglobin | F | | g/dL | 12.1 | 16.3 |
| 102 | Hematology | Lymphocytes | | | 10^9/L | 1 | 4.8 |
| 102 | Hematology | Monocytes | | | 10^9/L | 0.2 | 0.9 |

Page **44** of **61** 

| SITE | | | | | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | PANEL | <b>PARAMETER</b> | SEX | <b>AGE</b> | UNITS | LOW | HIGH |
| 102 | Hematology | Neutrophils | | | 10^9/L | 1.8 | 6.6 |
| 102 | Hematology | Platelet count | | | 10^9/L | 150 | 400 |
| 102 | Hematology | WBC count | | | 10^9/L | 4 | 11.1 |
| 102 | Urinalysis | Glucose | | | | NEGATIVE | |
| 102 | Urinalysis | Ketones | | | | NEGATIVE | |
| 102 | Urinalysis | Occult blood | | | | NEGATIVE | |
| 102 | Urinalysis | Protein | | | | NEGATIVE | |
| 102 | Urinalysis | Specific gravity | | | | 1.001 | 1.035 |
| 102 | Urinalysis | Urobilinogen | | | mg/dL | < 2.0 | |

 Table 10
 Site 103 Units and Reference Ranges by Parameter

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 103 | Chemistry | Albumin | | | g/dL | 3.4 | 5 |
| 103 | Chemistry | ALP | | | IU/L | 38 | 126 |
| 103 | Chemistry | ALT/SGPT | M | | IU/L | 17 | 63 |
| 103 | Chemistry | ALT/SGPT | F | | IU/L | 14 | 54 |
| 103 | Chemistry | AST/SGOT | | | IU/L | 15 | 41 |
| 103 | Chemistry | Bicarbonate | | | mmol/L | 21 | 31 |
| 103 | Chemistry | Blood urea nitrogen | | | mg/dL | 8 | 26 |
| 103 | Chemistry | Calcium | | | mg/dL | 8.4 | 10.2 |
| 103 | Chemistry | Chloride | | | mmol/L | 98 | 107 |
| 103 | Chemistry | Creatinine | | | mg/dL | 0.5 | 1.4 |
| 103 | Chemistry | Glucose | | | mg/dL | 65* | 95* |
| 103 | Chemistry | Magnesium | | | mg/dL | 1.6 | 2.3 |
| 103 | Chemistry | Phosphorous | | | mg/dL | 2.5 | 4.6 |
| 103 | Chemistry | Potassium | | | mmol/L | 3.5 | 5 |
| 103 | Chemistry | Sodium | | | mmol/L | 136 | 146 |
| 103 | Chemistry | Total Bilirubin | | | mg/dL | 0.3 | 1.5 |
| 103 | Chemistry | Total protein | | | g/dL | 6.3 | 7.7 |
| 103 | Hematology | Basophils | | | 10^9/L | 0 | 0.06 |
| 103 | Hematology | Eosinophils | | | 10^9/L | 0 | 0.4 |
| 103 | Hematology | Hematocrit | M | | % | 38 | 48.8 |
| 103 | Hematology | Hematocrit | F | | % | 34.1 | 43.3 |
| 103 | Hematology | Hemoglobin | M | | g/dL | 12.9 | 16.9 |
| 103 | Hematology | Hemoglobin | F | | g/dL | 11.6 | 14.6 |

| SITE | | | | | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | <b>PANEL</b> | <b>PARAMETER</b> | SEX | <b>AGE</b> | UNITS | LOW | HIGH |
| 103 | Hematology | Lymphocytes | | | 10^9/L | 0.8 | 3.65 |
| 103 | Hematology | Monocytes | | | 10^9/L | 0.3 | 0.9 |
| 103 | Hematology | Neutrophils | | | × 109/L | 1.42* | 6.34* |
| 103 | Hematology | Platelet count | | | × 109/L | 165* | 415* |
| 103 | Hematology | WBC count | | | 10^9/L | 3.8 | 10.6 |
| 103 | Urinalysis | Glucose | | | | Negative | |
| 103 | Urinalysis | Ketones | | | | Negative | |
| 103 | Urinalysis | Occult blood | | | | Negative | |
| 103 | Urinalysis | Protein | | | | Negative | |
| 103 | Urinalysis | Specific gravity | | | | 1.001 | 1.035 |
| 103 | Urinalysis | Urobilinogen | | | | Normal | |

 Table 11
 Site 104 Units and Reference Ranges by Parameter

| NUMBER PANEL PARAMETER SEX AGE UNITS LOW HIGH 104 Chemistry Albumin M g/dL 3.7 5.3 104 Chemistry Albumin F g/dL 4.2 5.5 104 Chemistry ALP U/L 34 104 104 Chemistry ALT/SGPT U/L 7 52 104 Chemistry AST/SGOT U/L 13 39 104 Chemistry Bicarbonate mmol/L 21 31 104 Chemistry Blood urea nitrogen mg/dL 7 25 104 Chemistry Calcium mg/dL 8.6 10.3 104 Chemistry Creatinine M mg/dL 98 107 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 85 125 104 | SITE | DANEI | DADAMETED | CEV | ACE | LIMITO | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|---|
| 104 Chemistry Albumin F g/dL 4.2 5.5 104 Chemistry ALP U/L 34 104 104 Chemistry ALT/SGPT U/L 7 52 104 Chemistry AST/SGOT U/L 13 39 104 Chemistry Bicarbonate mmol/L 21 31 104 Chemistry Blood urea nitrogen mg/dL 7 25 104 Chemistry Calcium mg/dL 8.6 10.3 104 Chemistry Chloride mmol/L 98 107 104 Chemistry Creatinine M mg/dL 0.7 1.3 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low-mg/dL 70 115 104 Chemistry Magnesium mg/dL 85 125 104 Chemistry Phosphorous | | | | | AGE | | | |
| 104 Chemistry ALT/SGPT U/L 7 52 104 Chemistry AST/SGOT U/L 13 39 104 Chemistry Bicarbonate mmol/L 21 31 104 Chemistry Blood urea nitrogen mg/dL 7 25 104 Chemistry Calcium mg/dL 8.6 10.3 104 Chemistry Chloride mmol/L 98 107 104 Chemistry Creatinine M mg/dL 0.7 1.3 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 70 115 104 Chemistry Glucose 51 - mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium | | | | F | | _ | | |
| 104 Chemistry AST/SGOT U/L 13 39 104 Chemistry Bicarbonate mmol/L 21 31 104 Chemistry Blood urea nitrogen mg/dL 7 25 104 Chemistry Calcium mg/dL 8.6 10.3 104 Chemistry Chloride mmol/L 98 107 104 Chemistry Creatinine M mg/dL 0.7 1.3 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 70 115 104 Chemistry Glucose 51 - mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium | 104 | Chemistry | ALP | | | U/L | 34 | 104 |
| 104 Chemistry Bicarbonate mmol/L 21 31 104 Chemistry Blood urea nitrogen mg/dL 7 25 104 Chemistry Calcium mg/dL 8.6 10.3 104 Chemistry Chloride mmol/L 98 107 104 Chemistry Creatinine M mg/dL 0.7 1.3 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 70 115 104 Chemistry Glucose 51 - mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin </th <th>104</th> <th>Chemistry</th> <th>ALT/SGPT</th> <th></th> <th></th> <th>U/L</th> <th>7</th> <th>52</th> | 104 | Chemistry | ALT/SGPT | | | U/L | 7 | 52 |
| 104 Chemistry nitrogen Blood urea nitrogen mg/dL 7 25 104 Chemistry Calcium mg/dL 8.6 10.3 104 Chemistry Chloride mmol/L 98 107 104 Chemistry Creatinine M mg/dL 0.7 1.3 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 70 115 104 Chemistry Glucose 51 - mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | AST/SGOT | | | U/L | 13 | 39 |
| 104 Chemistry Calcium mg/dL 8.6 10.3 104 Chemistry Chloride mmol/L 98 107 104 Chemistry Creatinine M mg/dL 0.7 1.3 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 70 115 50 50 mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Bicarbonate | | | mmol/L | 21 | 31 |
| 104 Chemistry Chloride mmol/L 98 107 104 Chemistry Creatinine M mg/dL 0.7 1.3 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 70 115 104 Chemistry Glucose 51 - mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | | | | mg/dL | 7 | 25 |
| 104 Chemistry Creatinine M mg/dL 0.7 1.3 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 70 115 104 Chemistry Glucose 51 - mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Calcium | | | mg/dL | 8.6 | 10.3 |
| 104 Chemistry Creatinine F mg/dL 0.6 1.2 104 Chemistry Glucose low - mg/dL 50 mg/dL mg/dL 70 115 104 Chemistry Glucose 51 - mg/dL high mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Chloride | | | mmol/L | 98 | 107 |
| 104 Chemistry Glucose low - mg/dL 50 70 115 104 Chemistry Glucose 51 - mg/dL 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Creatinine | M | | mg/dL | 0.7 | 1.3 |
| 104 Chemistry Glucose 51 - mg/dL high 85 125 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Creatinine | F | | mg/dL | 0.6 | 1.2 |
| high 104 Chemistry Magnesium mg/dL 1.9 2.7 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Glucose | | | mg/dL | 70 | 115 |
| 104 Chemistry Phosphorous mg/dL 2.5 5 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Glucose | | | mg/dL | 85 | 125 |
| 104 Chemistry Potassium mmol/L 3.5 5.1 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Magnesium | | | mg/dL | 1.9 | 2.7 |
| 104 Chemistry Sodium mmol/L 136 145 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Phosphorous | | | mg/dL | 2.5 | 5 |
| 104 Chemistry Total Bilirubin mg/dL 0 1.4 | 104 | Chemistry | Potassium | | | mmol/L | 3.5 | 5.1 |
| | 104 | Chemistry | Sodium | | | mmol/L | 136 | 145 |
| | 104 | Chemistry | Total Bilirubin | | | mg/dL | 0 | 1.4 |
| 104 Chemistry Total protein g/dL 6 8.3 | 104 | Chemistry | Total protein | | | g/dL | 6 | 8.3 |

| SITE | DANIEL | D. D. A. B. ETTED | CENT | . 65 | <b>TINITE</b> | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | LOW | HIGH |
| 104 | Hematology | Basophils | | | THOUS/MCL | 0 | 0.2 |
| 104 | Hematology | Eosinophils | | | THOUS/MCL | 0 | 0.5 |
| 104 | Hematology | Hematocrit | | | % | 39.5 | 50 |
| 104 | Hematology | Hemoglobin | | | g/dL | 13.5 | 16.9 |
| 104 | Hematology | Lymphocytes | | | THOUS/MCL | 0.9 | 3.3 |
| 104 | Hematology | Monocytes | | | THOUS/MCL | 0 | 0.8 |
| 104 | Hematology | Neutrophils | | | THOUS/MCL | 2 | 8.1 |
| 104 | Hematology | Platelet count | | | THOUS/MCL | 150 | 400 |
| 104 | Hematology | WBC count | | | THOUS/MCL | 4 | 10.5 |
| 104 | Urinalysis | Glucose | | | mg/dL | Negative | |
| 104 | Urinalysis | Ketones | | | mg/dL | Negative | |
| 104 | Urinalysis | Occult blood | | | /HPF | 2 | |
| 104 | Urinalysis | Protein | | | mg/dL | Negative | |
| 104 | Urinalysis | Specific gravity | | | | 1.003 | 1.03 |
| 104 | Urinalysis | Urobilinogen | | | mg/dL | < 2 | |

Table 12 Site 105 Units and Reference Ranges by Parameter

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 105 | Chemistry | Sodium | | | mEq/L | 135 | 145 |
| 105 | Chemistry | Potassium | | | mEq/L | 3.6 | 5.2 |
| 105 | Chemistry | Chloride | | | mEq/L | 98 | 108 |
| 105 | Chemistry | Bicarbonate | | | mEq/L | 22 | 32 |
| 105 | Chemistry | Calcium | | | mg/dL | 8.9 | 10.2 |
| 105 | Chemistry | Phosphorous | | | mg/dL | 2.5 | 4.5 |
| 105 | Chemistry | Magnesium | | | mg/dL | 1.8 | 2.4 |
| 105 | Chemistry | Blood urea<br>nitrogen | | | mg/dL | 8 | 21 |
| 105 | Chemistry | Albumin | | | g/dL | 3.5 | 5.2 |
| 105 | Chemistry | ALP | | | U/L | | |

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 105 | Chemistry | ALT/SGPT | M | 0 -<<br>50 | U/L | 10 | 64 |
| 105 | Chemistry | ALT/SGPT | M | 50 -<br>high | U/L | 10 | 48 |
| 105 | Chemistry | ALT/SGPT | F | | U/L | 7 | 33 |
| 105 | Chemistry | AST/SGOT | | | U/L | 9 | 38 |
| 105 | Chemistry | Creatinine | M | | mg/dL | 0.51 | 1.18 |
| 105 | Chemistry | Creatinine | F | | mg/dL | 0.38 | 1.02 |
| 105 | Chemistry | Glucose | | | mg/dL | 62 | 125 |
| 105 | Chemistry | Total Bilirubin | | | mg/dL | 0.2 | 1.3 |
| 105 | Chemistry | Total protein | | | g/dL | 6 | 8.2 |
| 105 | Hematology | Hematocrit | M | | % | 38 | 50 |
| 105 | Hematology | Hematocrit | F | | % | 36 | 45 |
| 105 | Hematology | Hemoglobin | M | | g/dL | 13 | 18 |
| 105 | Hematology | Hemoglobin | F | | g/dL | 11.5 | 15.5 |
| 105 | Hematology | Neutrophils | | | thou/uL | 1.8 | 7 |
| 105 | Hematology | Lymphocytes | | | thou/uL | 1 | 4.8 |
| 105 | Hematology | Monocytes | | | thou/uL | 0 | 0.8 |
| 105 | Hematology | Eosinophils | | | thou/uL | 0 | 0.5 |
| 105 | Hematology | Basophils | | | thou/uL | 1.8 | 7 |
| 105 | Hematology | Platelet count | | | thou/uL | 150 | 400 |
| 105 | Hematology | WBC count | | | x10^3/uL | 20 | 1000 |
| 105 | Urinalysis | Glucose | | | | Negative | |
| 105 | Urinalysis | Ketones | | | | Negative* | |
| 105 | Urinalysis | Occult blood | | | | 1.005 | 1.03 |
| 105 | Urinalysis | Protein | | | | negative | |
| 105 | Urinalysis | Specific gravity | | | | | |
| 105 | Urinalysis | Urobilinogen | | | | negative | |

 Table 13
 Site 107 Units and Reference Ranges by Parameter

| SITE | | | | | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| <b>NUMBER</b> | <b>PANEL</b> | <b>PARAMETER</b> | SEX | <b>AGE</b> | UNITS | LOW | HIGH |
| 107 | Chemistry | Albumin | | | g/L | 38 | 50 |
| 107 | Chemistry | ALP | | | U/L | 40 | 150 |
| 107 | Chemistry | ALT/SGPT | | | U/L | 7 | 40 |
| 107 | Chemistry | AST/SGOT | | | U/L | 5 | 34 |
| 107 | Chemistry | Bicarbonate | | | mmol/L | 23 | 29 |

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFER<br>HIC | |
|---|---|---|---|---|---|---|---|---|
| 107 | Chemistry | Blood urea<br>nitrogen | | | mmol/L | 2.5* | | 7.1* |
| 107 | Chemistry | Calcium | | | mmol/L | 2.2 | | 2.62 |
| 107 | Chemistry | Chloride | | | mmol/L | 100 | | 110 |
| 107 | Chemistry | Creatinine | M | | μmol/L | 64 | | 110 |
| 107 | Chemistry | Creatinine | F | | μmol/L | 50 | | 98 |
| 107 | Chemistry | Glucose | | | mmol/L | 3.8 | | 7 |
| 107 | Chemistry | Magnesium | | | mmol/L | 0.7 | | 1.1 |
| 107 | Chemistry | Phosphorous | | | mmol/L | 0.81* | | 1.4* |
| 107 | Chemistry | Potassium | | | mmol/L | 3.2 | | 5 |
| 107 | Chemistry | Sodium | | | mmol/L | 135 | | 145 |
| 107 | Chemistry | Total Bilirubin | | | μmol/L | low | < 23 | |
| 107 | Chemistry | Total protein | | | g/L | 65 | | 80 |
| 107 | Hematology | Hematocrit | | | L/L | 0.42 | | 0.54 |
| 107 | Hematology | Hematocrit | | | L/L | 0.33 | | 0.47 |
| 107 | Hematology | Hemoglobin | M | | g/L | 140 | | 180 |
| 107 | Hematology | Hemoglobin | F | | g/L | 120 | | 160 |
| 107 | Hematology | Neutrophils | | | 10^9/L | 2 | | 7.5 |
| 107 | Hematology | Lymphocytes | | | 10^9/L | 1.5 | | 4 |
| 107 | Hematology | Monocytes | | | 10^9/L | 0.2 | | 0.8 |
| 107 | Hematology | Eosinophils | | | 10^9/L | 0.04 | | 0.4 |
| 107 | Hematology | Basophils | | | 10^9/L | 0 | | 0.2 |
| 107 | Hematology | Platelet count | | | 10^9/L | 150 | | 400 |
| 107 | Hematology | WBC count | | | 10^9/L | 4 | | 11 |
| 107 | Urinalysis | Glucose | | | | Negative | | |
| 107 | Urinalysis | Ketones | | | | Negative | | |
| 107 | Urinalysis | Occult blood | | | | Negative | Trace | |
| 107 | Urinalysis | Protein | | | | Negative | Trace | |
| 107 | Urinalysis | Specific gravity | | | | 1.005 | | 1.03 |
| 107 | Urinalysis | Urobilinogen | | | umol/L | low | < 17 | |

Table 14 Site 110 Units and Reference Ranges by Parameter

| SITE | | | | - | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | <b>PANEL</b> | <b>PARAMETER</b> | SEX | <b>AGE</b> | UNITS | LOW | HIGH |
| 110 | Chemistry | Albumin | | | g/L | 39 | 50 |
| 110 | Chemistry | ALP | M | | U/L | 42 | 110 |
| 110 | Chemistry | ALP | F | | U/L | 32 | 93 |

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 110 | Chemistry | ALP | F | | U/L | 47 | 124 |
| 110 | Chemistry | ALT/SGPT | M | | U/L | 8 | 58 |
| 110 | Chemistry | ALT/SGPT | F | 16 -<br>50 | U/L | 7 | 36 |
| 110 | Chemistry | ALT/SGPT | F | 51 -<br>high | U/L | 8 | 45 |
| 110 | Chemistry | AST/SGOT | M | | U/L | 15 | 38 |
| 110 | Chemistry | AST/SGOT | F | 16 -<br>50 | U/L | 14 | 30 |
| 110 | Chemistry | AST/SGOT | F | 51 -<br>high | U/L | 15 | 37 |
| 110 | Chemistry | Bicarbonate | | | mmol/L | 21 | 31 |
| 110 | Chemistry | Blood urea nitrogen | M | 16 -<br>30 | mmol/L | 2.5 | 6.3 |
| 110 | Chemistry | Blood urea nitrogen | M | 31 -<br>40 | mmol/L | 3.1 | 8 |
| 110 | Chemistry | Blood urea nitrogen | M | 41 -<br>50 | mmol/L | 3.6 | 7.8 |
| 110 | Chemistry | Blood urea nitrogen | M | 50 -<br>high | mmol/L | 3 | 8.8 |
| 110 | Chemistry | Blood urea nitrogen | F | 16 -<br>40 | mmol/L | 2.5 | 6.4 |
| 110 | Chemistry | Blood urea nitrogen | F | 41 -<br>50 | mmol/L | 2.8 | 6.7 |
| 110 | Chemistry | Blood urea nitrogen | F | 50 -<br>high | mmol/L | 2.9 | 8 |
| 110 | Chemistry | Calcium | | 16 -<<br>59 | mmol/L | 2.11 | 2.55 |
| 110 | Chemistry | Calcium | | 59 -<br>high | mmol/L | 2.24 | 2.63 |
| 110 | Chemistry | Chloride | | | mmol/L | 100 | 109 |
| 110 | Chemistry | Creatinine | M | | umol/L | 67 | 109 |
| 110 | Chemistry | Creatinine | F | | umol/L | 49 | 882 |
| 110 | Chemistry | Glucose | | | mmol/L | 3.6* | 5.3* |
| 110 | Chemistry | Magnesium | | | mmol/L | 0.66 | 1.07 |
| 110 | Chemistry | Phosphorous | | | mmol/L | 0.88 | 1.45 |
| 110 | Chemistry | Potassium | | | mmol/L | 3.6 | 5 |
| 110 | Chemistry | Sodium | | | mmol/L | 136 | 148 |
| 110 | Chemistry | Total Bilirubin | | | umol/L | 4 | 23 |
| 110 | Chemistry | Total protein | | | g/L | 67 | 87 |
| 110 | Hematology | Hematocrit | M | | | 0.395 | 0.488 |
| 110 | Hematology | Hematocrit | F | | | 0.347 | 0.449 |

| SITE | | | ~=== | . ~= | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | LOW | HIGH |
| 110 | Hematology | Hemoglobin | M | | g/dL | 13.3 | 17.1 |
| 110 | Hematology | Hemoglobin | F | | g/dL | 11.5 | 14.8 |
| 110 | Hematology | Neutrophils | | | x10^9/L | 2.01 | 7.42 |
| 110 | Hematology | Lymphocytes | | | x10^9/L | 1.06 | 3.61 |
| 110 | Hematology | Monocytes | | | x10^9/L | 0.26 | 0.85 |
| 110 | Hematology | Eosinophils | | | x10^9/L | 0.02 | 0.45 |
| 110 | Hematology | Basophils | | | x10^9/L | 0.02 | 0.09 |
| 110 | Hematology | Platelet count | | | x10^9/L | 167 | 396 |
| 110 | Hematology | WBC count | | | x10^9/L | 3.89 | 9.93 |
| 110 | Urinalysis | Glucose | | | mg/dL | Negative | |
| 110 | Urinalysis | Ketones | | | mg/dL | Negative | |
| 110 | Urinalysis | Occult blood | | | | Negative | |
| 110 | Urinalysis | Protein | | | mg/dL | Negative | |
| 110 | Urinalysis | Specific gravity | | | | 1.005 | 1.03 |
| 110 | Urinalysis | Urobilinogen | | | E.U./dL | 0.2 | 1 |

 Table 15
 Site 111 Units and Reference Ranges by Parameter

| SITE | | | | | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | LOW | HIGH |
| 111 | Chemistry | Albumin | | | g/dL | 3.4 | 5 |
| 111 | Chemistry | ALP | | | U/L | 46 | 116 |
| 111 | Chemistry | ALT/SGPT | | | U/L | 12 | 78 |
| 111 | Chemistry | AST/SGOT | | | U/L | 15 | 37 |
| 111 | Chemistry | Bicarbonate | | | mEq/L | 21 | 32 |
| 111 | Chemistry | Blood urea nitrogen | | | mg/dL | 7 | 18 |
| 111 | Chemistry | Calcium | | | mg/dL | 8.5 | 10.4 |
| 111 | Chemistry | Chloride | | | mEq/L | 98 | 107 |
| 111 | Chemistry | Creatinine | | | mg/dL | 0.51 | 1.17 |
| 111 | Chemistry | Glucose | | | mg/dL | 70 | 110 |
| 111 | Chemistry | Magnesium | | | mg/dL | 1.8 | 2.4 |
| 111 | Chemistry | Phosphorous | | | mg/dL | 2.5 | 4.9 |
| 111 | Chemistry | Potassium | | | mEq/L | 3.5 | 5.1 |
| 111 | Chemistry | Sodium | | | mEq/L | 136 | 145 |
| 111 | Chemistry | Total Bilirubin | | | mg/dL | 0 | 1 |
| 111 | Chemistry | Total protein | | | g/dL | 6.4 | 8.2 |
| 111 | Hematology | Hematocrit | M | | % | 38 | 50 |

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 111 | Hematology | Hematocrit | F | AGE | % | 34 | 45 |
| 111 | Hematology | Hemoglobin | M | | g/dL | 13 | 17.5 |
| 111 | Hematology | Hemoglobin | F | | g/dL | 11.6 | 15.4 |
| 111 | Hematology | Neutrophils | | | K/uL | 1.5 | 8 |
| 111 | Hematology | Lymphocytes | | | K/uL | 1 | 4 |
| 111 | Hematology | Monocytes | | | K/uL | 0.2 | 1 |
| 111 | Hematology | Eosinophils | | | K/uL | 0 | 0.6 |
| 111 | Hematology | Basophils | | | K/uL | 0 | 0.2 |
| 111 | Hematology | Platelet count | | | K/uL | 140 | 390 |
| 111 | Hematology | WBC count | | | K/uL | 3.5 | 10.5 |
| 111 | Urinalysis | Glucose | | | | NEGATIVE | |
| 111 | Urinalysis | Ketones | | | | NEGATIVE | |
| 111 | Urinalysis | Occult blood | | | | NEGATIVE | |
| 111 | Urinalysis | Protein | | | mg/dL | < 10 | |
| 111 | Urinalysis | Specific gravity | | | | 1.005 | 1.035 |
| 111 | Urinalysis | Urobilinogen | | | EU/dL | 0.2 | 1 |

 Table 16
 Site 113 Units and Reference Ranges by Parameter

| SITE | | | - | , J | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | LOW | HIGH |
| 113 | Chemistry | Albumin | | Apr-<br>60 | g/dL | 3.4 | 4.2 |
| 113 | Chemistry | Albumin | | 61 -<br>70 | g/dL | 2.5 | 5.5 |
| 113 | Chemistry | Albumin | | 71 -<br>80 | g/dL | 3.6 | 4.8 |
| 113 | Chemistry | Albumin | | 81 -<br>90 | g/dL | 3.5 | 4.8 |
| 113 | Chemistry | Albumin | | 90 -<br>high | g/dL | 3.2 | 4.6 |
| 113 | Chemistry | ALP | | | IU/L | | |
| 113 | Chemistry | ALT/SGPT | M | | IU/L | 0 | 44 |
| 113 | Chemistry | ALT/SGPT | F | | IU/L | 0 | 32 |
| 113 | Chemistry | AST/SGOT | | | IU/L | 0 | 40 |
| 113 | Chemistry | Bicarbonate | | | mmol/L | 20 | 29 |
| 113 | Chemistry | Blood urea nitrogen | | 18 -<br>39 | mg/dL | 6 | 20 |
| 113 | Chemistry | Blood urea nitrogen | | 40 -<br>59 | mg/dL | 6 | 24 |
| 113 | Chemistry | Blood urea<br>nitrogen | | 60 -<br>89 | mg/dL | 8 | 27 |

Page **52** of **61** 

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 113 | Chemistry | Blood urea<br>nitrogen | SLIX | 90 -<br>high | mg/dL | 10 | |
| 113 | Chemistry | Calcium | | U | mg/dL | 4.5 | 5.6 |
| 113 | Chemistry | Chloride | | | mmol/L | 97 | 106 |
| 113 | Chemistry | Creatinine | | | mg/dL | 0.76 | 1.27 |
| 113 | Chemistry | Creatinine | | | mg/dL | 0.57 | 1 |
| 113 | Chemistry | Glucose | | | ng/mL | 65 | 199 |
| 113 | Chemistry | Magnesium | | | mg/dL | 1.6 | 2.3 |
| 113 | Chemistry | Phosphorous | | | mg/dL | 2.5 | 4.5 |
| 113 | Chemistry | Potassium | | | mmol/L | 3.5 | 5.2 |
| 113 | Chemistry | Sodium | | | mmol/L | 134 | 144 |
| 113 | Chemistry | Total Bilirubin | | | mg/dL | 0 | 1.2 |
| 113 | Chemistry | Total protein | | | g/dL | 6 | 8.5 |
| 113 | Hematology | Hematocrit | | | % | 43.5 | 53.7 |
| 113 | Hematology | Hemoglobin | | | g/dL | 14.1 | 18.1 |
| 113 | Hematology | Neutrophils | | | x10E3/uL | 1.4 | . 7 |
| 113 | Hematology | Lymphocytes | | | x10E3/uL | 0.7 | 3.1 |
| 113 | Hematology | Monocytes | | | x10E3/uL | 0.1 | 0.9 |
| 113 | Hematology | Eosinophils | | | x10E3/uL | 0 | 0.4 |
| 113 | Hematology | Basophils | | | x10E3/uL | 0 | 0.2 |
| 113 | Hematology | Platelet count | | | x10E3/uL | 150 | 450 |
| 113 | Hematology | WBC count | | | x10E3/uL | 3.4 | 10.8 |
| 113 | Urinalysis | Glucose | | | | Negative | |
| 113 | Urinalysis | Ketones | | | | Negative | |
| 113 | Urinalysis | Occult blood | | | | Negative | |
| 113 | Urinalysis | Protein | | | | Negative | |
| 113 | Urinalysis | Specific gravity | | | | 1 | 1.035 |
| 113 | Urinalysis | Urobilinogen | | | | Normal | |

Table 17 Site 116 Units and Reference Ranges by Parameter

| SITE | | | Ü | · | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | PANEL | <b>PARAMETER</b> | SEX | AGE | UNITS | LOW | HIGH |
| 116 | Chemistry | Albumin | | 20 -<br>60 | g/L | 35 | 52 |
| 116 | Chemistry | Albumin | | 61 -<br>90 | g/L | 32 | 46 |
| 116 | Chemistry | ALP | | | U/L | 40 | 150 |
| 116 | Chemistry | ALT/SGPT | | | U/L | < 56 | |

#### Rain Therapeutics Inc. RAIN-701 SAP

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 116 | Chemistry | AST/SGOT | | | U/L | 5 | 34 |
| 116 | Chemistry | Bicarbonate | | | mmol/L | 22 | 29 |
| 116 | Chemistry | Blood urea nitrogen | M | | mmol/L | 3.2 | 7.4 |
| 116 | Chemistry | Blood urea nitrogen | F | | mmol/L | 2.5 | 6.7 |
| 116 | Chemistry | Calcium | | | mmol/L | 2.1 | 2.55 |
| 116 | Chemistry | Chloride | | | mmol/L | 98 | 107 |
| 116 | Chemistry | Creatinine | M | | umol/L | 63.6 | 110.5 |
| 116 | Chemistry | Creatinine | F | | umol/L | 50.4 | 98.1 |
| 116 | Chemistry | Glucose | | | mmol/L | 3.6* | 5.3* |
| 116 | Chemistry | Magnesium | | | mmol/L | 0.66 | 1.07 |
| 116 | Chemistry | Phosphorous | | | mmol/L | 0.74 | 1.52 |
| 116 | Chemistry | Potassium | | | mmol/L | 3.5 | 5.1 |
| 116 | Chemistry | Sodium | | | mmol/L | 136 | 145 |
| 116 | Chemistry | Total Bilirubin | | | umol/L | 5.1 | 20.5 |
| 116 | Chemistry | Total protein | | | g/L | 64 | 83 |
| 116 | Hematology | Hematocrit | | M | % | 37 | 52 |
| 116 | Hematology | Hematocrit | | F | % | 35 | 47 |
| 116 | Hematology | Hemoglobin | | M | g/dL | 12.5 | 17.5 |
| 116 | Hematology | Hemoglobin | | F | g/dL | 11.5 | 16 |
| 116 | Hematology | Neutrophils | | | K/uL | 1.7 | 88 |
| 116 | Hematology | Lymphocytes | | | K/uL | 1 | 4.5 |
| 116 | Hematology | Monocytes | | | K/uL | 0.2 | 1 |
| 116 | Hematology | Eosinophils | | | K/uL | 0 | 0.5 |
| 116 | Hematology | Basophils | | | K/uL | 0 | 0.2 |
| 116 | Hematology | Platelet count | | | K/uL | 150 | 400 |
| 116 | Hematology | WBC count | | | × 109/L | 3.54* | 9.06* |
| 116 | Urinalysis | Glucose | | | | Negative | |
| 116 | Urinalysis | Ketones | | | | Negative | |
| 116 | Urinalysis | Occult blood | | | | Negative | |
| 116 | Urinalysis | Protein | | | | Negative | |
| 116 | Urinalysis | Specific gravity | | | | 1.001 | 1.035 |
| 116 | Urinalysis | Urobilinogen | | | | | |

 Table 18 Site 117 Units and Reference Ranges by Parameter

| SITE | | DADAMETED | C | · | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER<br>117 | PANEL Chemistry | PARAMETER<br>Albumin | SEX | <b>AGE</b> 18 - | g/dL | <b>LOW</b> 3.7 | HIGH 4.8 |
| 117 | Chemistry | Albuilliii | | 59 | g/uL | 3.7 | 4.0 |
| 117 | Chemistry | Albumin | | 60 -<br>89 | g/dL | 3.2 | 4.6 |
| 117 | Chemistry | Albumin | | 90 -<br>high | g/dL | 2.9 | 4.5 |
| 117 | Chemistry | ALP | | 15 -<br>20 | IU/L | 50 | 180 |
| 117 | Chemistry | ALP | | 20 -<br>high | IU/L | 40 | 140 |
| 117 | Chemistry | ALT/SGPT | | | | 7* | 41* |
| 117 | Chemistry | AST/SGOT | | | | 12* | 38* |
| 117 | Chemistry | Bicarbonate | | | meq/L | 22* | 30* |
| 117 | Chemistry | Blood urea nitrogen | | | mg/dL | 10 | 25 |
| 117 | Chemistry | Calcium | | | mg/dL | 8.6 | 10.4 |
| 117 | Chemistry | Chloride | | | mmol/L | 98 | 111 |
| 117 | Chemistry | Creatinine | M | | mg/dL | < 1.28 | |
| 117 | Chemistry | Creatinine | F | | mg/dL | < 1.16 | |
| 117 | Chemistry | Glucose | | | mg/dL | 50 | 140 |
| 117 | Chemistry | Magnesium | | | mg/dL | 1.8 | 2.3 |
| 117 | Chemistry | Phosphorous | | | mg/dL | 2.5 | 4.5 |
| 117 | Chemistry | Potassium | | | mmol/L | 3.5 | 5 |
| 117 | Chemistry | Sodium | | | mmol/L | 135 | 145 |
| 117 | Chemistry | Total Bilirubin | | | mg/dL | < 1.2 | |
| 117 | Chemistry | Total protein | | | g/dL | 6 | 8.3 |
| 117 | Hematology | Hematocrit | M | | % | 41 | 53 |
| 117 | Hematology | Hematocrit | F | | % | 36 | 46 |
| 117 | Hematology | Hemoglobin | M | | g/dL | 13.5 | 17 |
| 117 | Hematology | Hemoglobin | F | | g/dL | 12 | 15 |
| 117 | Hematology | Neutrophils | | | K/uL | 1.8 | 7.7 |
| 117 | Hematology | Lymphocytes | | | K/uL | 1.1 | 4 |
| 117 | Hematology | Monocytes | | | K/uL | 0 | 0.8 |
| 117 | Hematology | Eosinophils | | | K/uL | 0 | 0.7 |
| 117 | Hematology | Basophils | | | K/uL | 0 | 0.2 |
| 117 | Hematology | Platelet count | | | K/uL | 150 | 450 |
| 117 | Hematology | WBC count | | | K/uL | 3.8 | 10.6 |

| SITE | | | | | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | <b>PANEL</b> | <b>PARAMETER</b> | SEX | <b>AGE</b> | UNITS | LOW | HIGH |
| 117 | Urinalysis | Glucose | | | | Negative | |
| 117 | Urinalysis | Ketones | | | | Negative | |
| 117 | Urinalysis | Occult blood | | | | Negative | |
| 117 | Urinalysis | Protein | | | | Negative | |
| 117 | Urinalysis | Specific gravity | | | | 1.005 | 1.03 |
| 117 | Urinalysis | Urobilinogen | | | U/dL | < 2.0 | |

**Table 19 Site 122 Units and Reference Ranges by Parameter** 

| SITE<br>NUMBER | PANEL | PARAMETER | SEX | | UNITS | REFERENCE<br>LOW | REFERENCE<br>HIGH |
|---|---|---|---|---|---|---|---|
| 122 | Chemistry | Albumin | | | g/dL | 3.5 | 5.2 |
| 122 | Chemistry | ALP | M | | U/L | 40 | 130 |
| 122 | Chemistry | ALP | F | | U/L | 35 | 105 |
| 122 | Chemistry | ALT/SGPT | M | | U/L | low | 41 |
| 122 | Chemistry | ALT/SGPT | F | | U/L | low | 33 |
| 122 | Chemistry | AST/SGOT | M | | U/L | low | 40 |
| 122 | Chemistry | AST/SGOT | F | | U/L | low | 32 |
| 122 | Chemistry | Bicarbonate | | | meq/L | 22* | 30* |
| 122 | Chemistry | Blood urea nitrogen | | 18 -<<br>60 | mg/dL | 6 | 20 |
| 122 | Chemistry | Blood urea nitrogen | | 60 -<br>90 | mg/dL | 8 | 23 |
| 122 | Chemistry | Blood urea nitrogen | | > 90 | mg/dL | 8.6 | 10 |
| 122 | Chemistry | Calcium | | 18 -<<br>60 | mg/dL | 8.6 | 10 |
| 122 | Chemistry | Calcium | | 60 -<br>90 | mg/dL | 8.8 | 10.2 |
| 122 | Chemistry | Calcium | | > 90 | mg/dL | 8.2 | 9.6 |
| 122 | Chemistry | Chloride | | | mmol/L | 98 | 107 |
| 122 | Chemistry | Creatinine | M | | mg/dL | 0.7 | 1.2 |
| 122 | Chemistry | Creatinine | F | | mg/dL | 0.5 | 0.9 |
| 122 | Chemistry | Glucose | | | mg/dL | 74 | 109 |
| 122 | Chemistry | Magnesium | | 20 -<<br>60 | mg/dL | 1.6 | 2.6 |
| 122 | Chemistry | Magnesium | | 60 -<br>90 | mg/dL | 1.6 | 2.4 |
| 122 | Chemistry | Phosphorous | | | mg/dL | 2.5 | 4.5 |
| 122 | Chemistry | Potassium | | | mmol/L | 3.4 | 4.5 |
| 122 | Chemistry | Sodium | | | mmol/L | 136 | 145 |

#### Rain Therapeutics Inc. RAIN-701 SAP

| SITE | | | | | | REFERENCE | REFERENCE |
|---|---|---|---|---|---|---|---|
| NUMBER | PANEL | PARAMETER | SEX | AGE | UNITS | LOW | HIGH |
| 122 | Chemistry | Total Bilirubin | | | mg/dL | low | 1.2 |
| 122 | Chemistry | Total protein | | | g/dL | 6.4 | 8.3 |
| 122 | Hematology | Hematocrit | M | | % | 40.1 | 51 |
| 122 | Hematology | Hematocrit | F | | % | 34.1 | 44.9 |
| 122 | Hematology | Hemoglobin | M | | g/dL | 13.7 | 17.5 |
| 122 | Hematology | Hemoglobin | F | | g/dL | 11.2 | 15.7 |
| 122 | Hematology | Neutrophils | | | k/uL | 2.3 | 7.1 |
| 122 | Hematology | Lymphocytes | | | k/uL | 0.8 | 3.5 |
| 122 | Hematology | Monocytes | | | k/uL | 0.2 | 0.8 |
| 122 | Hematology | Eosinophils | | | k/uL | 0.1 | 0.4 |
| 122 | Hematology | Basophils | | | k/uL | 0 | 0.1 |
| 122 | Hematology | Platelet count | | | k/uL | 150 | 450 |
| 122 | Hematology | WBC count | | | k/uL | 4 | 10.5 |
| 122 | Urinalysis | Glucose | | | | Negative | |
| 122 | Urinalysis | Ketones | | | | Negative | |
| 122 | Urinalysis | Occult blood | | | | Negative | |
| 122 | Urinalysis | Protein | | | | Negative | |
| 122 | Urinalysis | Specific gravity | | | | 1.001 | 1.03 |
| 122 | Urinalysis | Urobilinogen | | | | Normal | |


Rain Therapeutics Inc. RAIN-701 SAP

# 18 Appendix B: Common Terminology Criteria for Adverse Events for Laboratory Parameters

Table 20 Common Terminology Criteria for Adverse Events v5.0. November 27, 2017

| Laur | | | Table 20 Common telliminology efficial for Adverse Events 43.6, 100 cm feet, 2017 | LS V J.U9 LIUV VIIIR | 107 6/7 10 | | | |
|---|---|---|---|---|---|---|---|---|
| Panel | Parameter | CTCAE Term | Definition | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Chemistry | Sodium | Hypernatremia | A disorder characterized by laboratory test results that indicate an elevation in the concentration of sodium in the blood. | >ULN - 150<br>mmol/L | >150 - 155 mmol/L; intervention initiated | >155 - 160<br>mmol/L;<br>hospitalization<br>indicated | >160 mmol/L;<br>life-threatening<br>consequences | Death |
| Chemistry | Sodium | Hyponatremia | A disorder characterized by laboratory test results that indicate a low concentration of sodium in the blood. | <pre><lln -="" 130="" l<="" mmol="" pre=""></lln></pre> | 125-129 mmol/L and asymptomatic | 125-129 mmol/L<br>symptomatic; 120-<br>124 mmol/L<br>regardless of<br>symptoms | <120 mmol/L; life-threatening consequences | Death |
| Chemistry | Potassium | Hyperkalemia | A disorder characterized by laboratory test results that indicate an elevation in the concentration of potassium in the blood; associated with kidney failure or sometimes with the use of diuretic drugs | >ULN - 5.5<br>mmol/L | >5.5 - 6.0 mmol/L;<br>intervention<br>initiated | >6.0 - 7.0 mmol/L;<br>hospitalization<br>indicated | >7.0 mmol/L; life-<br>threatening<br>consequences | Death |
| Chemistry | Potassium | Hypokalemia | A disorder characterized by laboratory test results that indicate a low concentration of potassium in the blood. | <lln -="" 3.0<br="">mmol/L</lln> | Symptomatic with <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" th=""><th>&lt;3.0 - 2.5 mmoVL;<br/>hospitalization<br/>indicated</th><th>&lt;2.5 mmol/L; life-<br/>threatening<br/>consequences</th><th>Death</th></lln> | <3.0 - 2.5 mmoVL;<br>hospitalization<br>indicated | <2.5 mmol/L; life-<br>threatening<br>consequences | Death |
| Chemistry | Calcium | Hyper-calcemia | A disorder characterized by laboratory test results that indicate an elevation in the concentration of calcium (corrected for albumin) in blood. | >ULN - 2.9<br>mmol/L | >2.9 - 3.1 mmol/L;<br>symptomatic | >3.1 - 3.4 mmol/L;<br>hospitalization<br>indicated | >3.4 mmol/L; life-<br>threatening<br>consequences | Death |
| Chemistry | Calcium | Hypocalcemia | A disorder characterized by laboratory test results that indicate a low concentration of calcium (corrected for albumin) in the blood. | <lln -="" 2.0<br="">mmol/L</lln> | <2.0 - 1.75 mmol/L; symptomatic | <pre>&lt;1.75 - 1.5 mmo//L; hospitalization indicated</pre> | <1.5 mmol/L; life-<br>threatening<br>consequences | Death |

# Rain Therapeutics Inc. RAIN-701 SAP

| Grade 4 Grade 5 | | | | <pre></pre> <pre>&lt;</pre> | <pre>consequences &lt;0.7 mg/dL; &lt;0.3 mmol/L; lifethreatening consequences &lt;30 mg/dL; &lt;1.7 mmol/L; lifethreatening consequences; seizures &gt;6.0 x ULN</pre> | consequences <ul> <li>co.7 mg/dL; &lt;0.3 mmol/L;</li> <li>lifethreatening consequences</li> <li>consequences;</li> <li>consequences;</li> <li>seizures</li> <li>&gt;6.0 x ULN if baseline was normal; &gt;10.0 x baseline if baseline was abnormal</li> </ul> |
|---|---|---|---|---|---|---|
| | | | | 1 11 11 11 | ٠ | |
| >3.0 - 8.0 mg/dL;<br>>1.23 - 3.30<br>mmol/L | | <0.9 - 0.7 mg/dL;<br><0.4 - 0.3 mmol/L | <pre>&lt;40 - 30 mg/dL;<br/>&lt;2.2 - 1.7 mmol/L</pre> | | >3.0 x baseline;<br>>3.0 - 6.0 x ULN | |
| | | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <55 - 40 mg/dL;<br><3.0 - 2.2 mmol/L | | >1.5 - 3.0 x<br>baseline; >1.5 -<br>3.0 x ULN | >1.5 - 3.0 x<br>baseline; >1.5 -<br>3.0 x ULN<br>>1.5 - 3.0 x ULN<br>if baseline was<br>normal; >1.5 - 3.0<br>x baseline if<br>baseline was<br>abnormal |
| Grade 1 Grade 2 | >ULN - 3.0<br>mg/dL; >ULN -<br>1.23 mmol/L | <pre><lln -="" 0.5="" 1.2="" <lln="" dl;="" l<="" mg="" mmol="" pre=""></lln></pre> | <pre><lln -="" 3.0="" 55="" <lln="" dl;="" l<="" mg="" mmol="" pre=""></lln></pre> | | >ULN - 1.5 x > ULN - 1.5 x b | ne<br>1.0 |
| Deliminon | A disorder characterized by laboratory test results that indicate an elevation in the concentration of magnesium in the blood. | A disorder characterized by laboratory test results that indicate a low concentration of magnesium in the blood. | A disorder characterized by laboratory test results that indicate a low concentration of glucose in | the blood. | the blood. A finding based on laboratory test results that indicate increased levels of creatinine in a biological specimen. | A finding based on laboratory test results that indicate increased levels of creatinine in a biological specimen. A finding based on laboratory test results that indicate an abnormally high level of bilirubin in the blood. Excess bilirubin is associated with jaundice. |
| | Hypermagnesemia | Hypomagnesemia | Hypoglycemia | | Creatinine | Creatinine<br>increased<br>Blood bilirubin<br>increased |
| Parameter | Magnesium | Magnesium | Glucose | | Creatinine | Creatinine<br>Total<br>Bilirubin |
| Panel | Chemistry | Chemistry | Chemistry | | Chemistry | Chemistry |

# Version 1.0, 14 October 2022

## Rain Therapeutics Inc. RAIN-701 SAP

| Parameter | CTCAE Term | Definition | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| ALT/SGPT | Alanine<br>aminotransferase<br>increased | A finding based on laboratory test results that indicate an increase in the level of alanine aminotransferase (ALT or SGPT) in the blood specimen. | >ULN if baseline<br>was normal; 1.5 -<br>3.0 x baseline if<br>baseline was<br>abnormal | >3.0 - 5.0 x ULN if baseline was normal; >3.0 - 5.0 x baseline if baseline was abnormal | if baseline was<br>normal; >5.0 - 20.0 x ULN<br>if baseline was<br>normal; >5.0 -<br>20.0 x baseline if<br>baseline was<br>abnormal | >20.0 x ULN if<br>baseline was<br>normal; >20.0 x<br>baseline if baseline<br>was abnormal | |
| ALP | Alkaline<br>phosphatase<br>increased | A finding based on laboratory test results that indicate an increase in the level of alkaline phosphatase in a blood specimen. | >ULN - 2.5 x<br>ULN if baseline<br>was normal; 2.0 -<br>2.5 x baseline if<br>baseline was<br>abnormal | >2.5 - 5.0 x ULN if baseline was normal; >2.5 - 5.0 x baseline if baseline was abnormal | >5.0 - 20.0 x ULN if baseline was normal; >5.0 - 20.0 x baseline if baseline was abnormal | >20.0 x ULN if<br>baseline was<br>normal; >20.0 x<br>baseline if baseline<br>was abnormal | |
| Albumin | Hypoalbuminemia | A disorder characterized by laboratory test results that indicate a low concentration of albumin in the blood. | <lln -="" 3="" 30="" dl;<="" g="" l<="" ln="" th=""><th>&lt;3 - 2 g/dL; &lt;30 -<br/>20 g/L</th><th>&lt;2 g/dL; &lt;20 g/L</th><th>Life-threatening consequences; urgent intervention indicated</th><th>Death</th></lln> | <3 - 2 g/dL; <30 -<br>20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences; urgent intervention indicated | Death |
| Hemoglobin | Anemia | A disorder characterized by a reduction in the amount of hemoglobin in 100 ml of blood. Signs and symptoms of anemia may include pallor of the skin and nucous membranes, shortness of breath, palpitations of the heart, soft systolic murmurs, lethargy, and fatigability. | <pre><lln -="" 10.0="" 100="" 6.2="" <lln="" dl;="" g="" l;="" l<="" mmol="" pre=""></lln></pre> | <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | <pre>&lt;8.0 g/dL; &lt;4.9 mmol/L; &lt;80 g/L; transfusion indicated</pre> | Life-threatening<br>consequences;<br>urgent intervention<br>indicated | Death |
| Hemoglobin | Hemoglobin<br>increased | A finding based on laboratory test results that indicate increased levels of hemoglobin above normal. | Increase in >0 - 2<br>g/dL | Increase in >2 - 4<br>g/dL | Increase in >4<br>g/dL | | |
| Neutrophils | Neutrophil count<br>decreased | A finding based on laboratory test results that indicate a decrease in number of neutrophils in a blood specimen. | <pre><lln -="" 1.5x="" 10e9="" 1500="" <lln="" l<="" mm3;="" pre=""></lln></pre> | <1500 -<br>1000/mm3; <1.5 -<br>1.0x 10e9 /L | <1000 - 500/mm3;<br><1.0 - 0.5 x10e9<br>/L | <500/mm3; <0.5 x<br>10e9 /L | |

# Rain Therapeutics Inc. RAIN-701 SAP

| Panel | Parameter | CTCAE Term Definition | Definition | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|---|
| Hematology | Hematology Lymphocytes | Lymphocyte count<br>decreased | A finding based on laboratory test results that indicate a decrease in number of lymphocytes in a blood specimen. | <lln -="" 800="" mm3;<br=""><lln -="" 0.8="" x<br="">10e9/L</lln></lln> | <800 - 500/mm3;<br><0.8 - 0.5 x<br>10e9/L | <500 - 200/mm3;<br><0.5 - 0.2 x<br>10e9/L | <200/mm3; <0.2 x<br>10e9/L | |
| Hematology | Eosinophils | Eosinophilia | A disorder characterized by laboratory test results that indicate an increased number of eosinophils in the blood. | >ULN and >Baseline | | Steroids initiated | | |
| Hematology | Platelet<br>count | Platelet count<br>decreased | A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen. | <lln -="" 75.0="" x<br="">10e9/L</lln> | <75.0 - 50.0 x<br>10e9/L | <50.0 - 25.0 x<br>10e9/L | <25.0 x 10e9/L | |